# "Effect of Physical Therapy on NLRP3 Inflammasome Activation and Muscle Atrophy in Critical Illness Myopathy"

Óscar Leonardo Arellano Pérez

Doctoral Thesis Project Submitted in Candidacy for the Degree of Doctor in Biomedical Sciences

Aug 11, 2025

# **Table of Contents**

| Αl | bstract | | . 4 |
|---|---|---|---|
| 1. | Back | groundground | . 5 |
| | 1.1. | Critical illness myopathy | . 5 |
| | 1.2. | Potential Mechanisms and Pathogenesis of CIM | . 6 |
| | 1.3. | Muscle Atrophy, Inflammation, and the NLRP3 Inflammasome | . 6 |
| | 1.4. | NLRP3 Inflammasome Activation in CIM: Priming and Oligomerization | |
| | 1.5. | Physical Therapy, Inflammation, and Potential Modulation of the NLRP3 Inflammasom | e |
| | in CIM | 8 | |
| 2. | Нурс | othesis | . 9 |
| 3. | Gene | neral Objective | |
| 4. | Spec | ific Objectives | . 9 |
| 5. | Expe | rimental Design | 10 |
| 6. | Patie | ents and Methods | 12 |
| | 6.1. | Study Design | 12 |
| | 6.2. | Patients | 12 |
| | 6.2.1 | | |
| | 6.2.2 | , , , | |
| | 6.2.3 | | |
| | 6.3. | Sample Size Validation | |
| | 6.4. | Sample Collection from Patients with CIM and Controls | |
| | 6.4.1 | 1 / | |
| | 6.4.2 | Blood Samples | 13 |
| | 6.5. | Evaluators | 13 |
| | 6.6. | Histological and Biochemical Methods | |
| | 6.6.1 | | |
| | 6.6.2.<br>6.6.3. | | |
| | 6.6.4 | | |
| | 6.6.5 | • | |
| | 6.6.6 | Microarray | 16 |
| | 6.7. | Demographic Variables, Severity of Critical Illness, Clinical Assessment of Muscle | |
| | • | h, and Functionality | |
| _ | 6.8. | Statistical Analysis | |
| 7. | | al Considerations | |
| | 7.1. | Social Utility | |
| | 7.2. | Protection of Vulnerable Groups | |
| | 7.3. | Randomization | 18 |
| | 7.4. | Adverse Events | 19 |
| | 7.5. | Benefit Assessment | 19 |
| | 7.6. | Protection of Privacy | 20 |
| | 7.7. | Ethical Monitoring of the Project | 20 |

| 7.8. Feasibility | 20 |
|---------------------------------------------|----|
| 8. Discussion | 21 |
| 10. Gantt Chart | 32 |
| Appendix 2. Ultrasound Evaluation Procedure | 33 |

#### Abstract

Critical Illness myopathy (CIM) is a common cause of acquired weakness in the intensive care unit. It is defined as a proximal predominant tetra-paresis, usually symmetrical and with respiratory muscle involvement. This condition is a usual complication in intensive care unit (ICU) and has been associated with increased mortality and healthcare costs. Myopathy in the critically ill patient can progress to post-intensive care syndrome, which results in persistent cognitive, mental and physical dysfunction. In Chile, 40% of patients with critical illness due to COVID-19 developed this syndrome. This pathology presents muscle atrophy and alters of contractility, and several cellular mechanisms have been associated with its development, but its etiopathogenesis is still unclear. The role of the ubiquitin proteosome system and atrogenes expression has been linked to its genesis. In murine models of sepsis and denervation, which replicate the characteristics of the critically ill patient. NLRP3 inflammasome complex produces muscle atrophy by overexpression of atrogenes. The NLRP3 inflammasome is a multiprotein complex that plays a pivotal role in inflammatory signalling, and secretion of IL-1β and IL-18. Overexpression of this complex has been reported in CIM, but is NLRP3 inflammasome activation associated with muscle atrophy due to atrogen upregulation in critically ill patients? One of the most important risk factors for this myopathy is mechanical silencing, which, unlike other factors, is modifiable by early mobilization. Physical therapy has demonstrated different effects at the cellular level in the skeletal muscle of these patients. In different pathological conditions, physical therapy is a regulator of inflammation, IL-1β and NLRP3 inflammasome levels, but does physical therapy decrease NLRP3 inflammasome activation in the skeletal muscle of patients with CPM, ¿thereby contributing to a reduction in muscle atrophy? Based on this background, the following hypothesis is proposed: Physical therapy decreases NLRP3 inflammasome activity and reduces muscle atrophy in critical illness myopathy. To test this assertion, in the early stage of ICU stay, patients at risk of this condition (n=16) will be randomized to be treated with conventional physical therapy or to additional physical therapy using servo-assisted motorized movement therapy device, 2 times a day for 60 minutes. In addition, patients without this condition will be considered as controls (n=8). From biopsy samples of the vastus lateralis muscle, histology studies will be performed to determine muscle atrophy and the structure of cellular organelles, expression of atrogenes mRNA by RT-qPCR, protein levels of key mediators involved with NLRP3 inflammasome activation by Western blot, and transcriptomics by microarray. The above to address the following specific aims: a) To evaluate the effect of physical therapy on NLRP3 inflammasome activation in vastus lateralis biopsies from patients with CIM, and to compare this activity with control patients, b) To evaluate the effect of physical therapy on muscle atrophy in vastus lateralis biopsies from patients with CIM, and to relate these results with NLRP3 inflammasome activation, c) To evaluate the effect of physical therapy on the gene expression profile of signalling pathways involved in skeletal muscle atrophy in patients with CIM, and d) To analyze the association between gene expression and skeletal muscle biochemical parameters with the clinical diagnosis of CIM. Extra physical therapy is expected to decrease NLRP3 inflammasome activation, muscle atrophy, and differential expression of genes related to the development of CIM. Additionally, it is expected that these variables are associated with the clinical and ultrasound diagnosis of CIM. **Due to** the functional deficit suffered by patients who survive critical illness, it is importance to study the mechanisms underlying to this disorder. This study proposes a translational approach to achieve this purpose, furthermore, to explore the contribution of the nonpharmacological intervention for the prevention and management of the critical illness myopathy: the physical therapy.

# 1. Background

# 1.1.Critical illness myopathy

Critical illness myopathy is a common cause of intensive care unit-acquired weakness (ICUAW)(1). ICUAW is a neuropathy and/or myopathy characterized by symmetric, predominantly proximal muscle weakness(2,3), without involvement of facial or ocular muscles(3,4). Respiratory muscles may also be affected(4,5), leading to diaphragmatic dysfunction associated with mechanical ventilation (ventilator-induced diaphragmatic dysfunction, VIDD), which complicates weaning from ventilatory support(6). ICU-AW may be triggered by: a) a neurogenic disorder known as critical illness polyneuropathy (CIP), b) a myogenic disorder referred to as critical illness myopathy (CIM), and/or c) the coexistence of both conditions (4.7-10). CIP is an acute, acquired sensorimotor axonal neuropathy caused by inflammation of the peripheral nerves (6,11). CIM is characterized by impaired muscle mass and contractility<sup>6,12</sup>, and presents with pathognomonic signs such as preserved sensory function, elevated creatine kinase levels(11), and most notably, a preferential loss of myosin compared to actin in muscle biopsy samples(6,12,13). Since muscle atrophy and impaired contractility are key features associated with increased mortality(14-18) and physical disability(19.20), much of the research has focused on CIM and the molecular pathways involved in skeletal muscle degradation(21).

The development of critical illness myopathy (CIM) is associated with the severity of the critical illness(22-24). Both modifiable and non-modifiable risk factors have been identified(3,4,25). Modifiable factors include hyperglycaemia(8,25–28), parenteral nutrition(4,8,25,27,29), use of agents(4,25,27), neuromuscular blockade(4,8,10,11,25,27,28,30,31), vasopressor corticosteroid therapy(2,4,8,11,25,27,31), prolonged sedation and analgesia(4,25,31), use of aminoglycoside antibiotics(4,25,26,28), prolonged mechanical ventilation(2,8,25-27,29,31), extended ICU stay(8,29), and mechanical silencing due to prolonged immobilization(4,25,27-29,31). Non-modifiable risk factors include specific diagnoses and life-support measures associated with critical illness, such as sepsis(25-27,29,32), systemic inflammatory response syndrome (SIRS)(4,8,25,32), multiple organ failure (MOF)(2,4,25-27,32), hyperlactatemia(4), and renal replacement therapy(26). Patient-related characteristics such as age(4,25,29), comorbidities(4), and female sex (4,25,27) have also been identified as non-modifiable contributors.

Regarding the diagnosis of CIM, different strategies are employed depending on whether the patient is cooperative or non-cooperative. Another key aspect is the differential diagnosis between CIM and CIP. In awake and cooperative patients, muscle strength is clinically assessed using the Medical Research Council Sum Score (MRC-SS)(3,9,33). A score of 48 or below indicates muscle weakness, with scores below 36 denoting severe weakness (4,33,34). Handgrip dynamometry is another diagnostic tool in conscious patients; values below 11 kg for men and 7 kg for women are indicative of CIM. However, the validity of handgrip strength as a representative measure of global muscle strength has been questioned (35). Electrophysiological evaluation is also used to diagnose CIM and can be applied in unconscious or non-cooperative patients, as well as for differential diagnosis between CIP and CIM(34.36). Nerve and muscle biopsies may provide valuable mechanistic insight and enable differential diagnosis; however, due to their invasive nature, biopsies are recommended only within a research context(33,34). In non-cooperative patients, various imaging techniques have been employed to assess muscle mass as a surrogate for muscle strength. Computed tomography (CT) and magnetic resonance imaging (MRI) allow for the evaluation of muscle quality, detection of fatty infiltration, and quantification of lean muscle mass(16); Nevertheless, these methods are costly and require specialized personnel and software (16,34). Among imaging tools, quadriceps muscle ultrasound appears the most promising, as it permits rapid, bedside, and repeatable assessments of both quantitative parameters (muscle thickness. anatomical and physiological cross-sectional area) and qualitative features (echogenicity and muscle architecture)(18,34,37). Diagnosis of CIM by muscle ultrasound is based on changes in sonographic variables observed within 7 to 10 days of critical illness progression, including a ≥20% reduction in muscle thickness, ≥10% decrease in cross-sectional area, ≥5% decrease in pennation angle, and an 8-10% increase in echogenicity (17,18,37). Early diagnosis is of critical importance, as protein degradation, muscle mass loss (38,39), and electrophysiological alterations(40) occur within the first 10 days of ICU admission. iven the relevance of early detection, several critical illness severity scores—such as the Sequential Organ Failure Assessment (SOFA) and the Acute Physiology and Chronic Health Evaluation II (APACHE II)—have been proposed. When combined with muscle ultrasound assessment, these tools may be sufficient to raise suspicion and support the clinical consideration of this condition (22,23,41,42).

CIM is a common complication among critically ill patients (17,31,43) and is associated with increased mortality (9,11,25,28,29,31), prolonged hospital stays (9,10,25,28), longer durations of mechanical ventilation (10,29), higher healthcare costs, and reduced long-term physical function and quality of life (9,10,29,31,44). Moreover, this condition may progress to post-intensive care syndrome (PICS), which can result in persistent cognitive, mental, and physical dysfunction (4,28,45). A multicentre Chilean study evaluating the functional and cognitive sequelae of PICS in patients who experienced critical illness due to COVID-19 found that 40% of survivors exhibited some degree of disability after hospital discharge (46). Therefore, understanding the cellular and molecular etiopathogenesis of CIM is essential for developing both pharmacological and non-pharmacological therapeutic strategies.

# 1.2. Potential Mechanisms and Pathogenesis of CIM

CIM is characterized by reduced muscle mass and impaired contractility(44,47–49). In vivo muscle biopsies from critically ill patients, postmortem tissue samples, and animal models of CIM have revealed skeletal muscle fiber atrophy and degeneration(21,50–52). Biopsies from patients with CIM suggest that these alterations result from an imbalance between protein synthesis and degradation, the latter being exacerbated through: a) activation of the ubiquitin-proteasome system (UPS), b) cytosolic proteases such as calpains and caspases, and c) dysregulation of autophagy pathways. Additional mechanisms described include decreased muscle excitability, impaired neuromuscular transmission, channelopathies, altered calcium homeostasis, mitochondrial dysfunction, and oxidative stress, among others(4,33,38,44,53). Although multiple etiological mechanisms have been proposed in the pathophysiology of CIM, its precise aetiology and causative pathways remain unclear. Therefore, further biomedical research is needed to elucidate the pathogenesis of CIM and to develop novel preventive and therapeutic strategies.

# 1.3. Muscle Atrophy, Inflammation, and the NLRP3 Inflammasome

The primary risk factors for the loss of muscle mass and strength, hallmarks of CIM, include sepsis, SIRS, and elevated levels of inflammatory markers (54). Among the proinflammatory cytokines involved in the development of muscle atrophy are tumor necrosis factor-alpha (TNFα), interleukin-6 (IL-6), and interleukin-1 (IL-1)(55). In addition to systemic inflammation, skeletal muscle is now recognized as a secretory organ capable of releasing various myokines (peptides, metabolites, cytokines, among others), including IL-6 and IL-1\(\textit{B}\). (55). The processes of gene expression, cleavage, and secretion of IL-1β are tightly regulated(56). Since IL-1β is translated as an inactive precursor (pro-IL-1β), its cleavage is mediated by the NLRP3 inflammasome (55,56), a multiprotein complex essential to inflammatory signalling (57). This complex is composed of the NLRP3 receptor protein, the ASC adaptor protein, and procaspase-1 as the effector component(57). In addition to its role as a key regulator of muscle metabolism(58,59), the NLRP3 inflammasome has been implicated in various myopathies(60-62), the development of sarcopenia(63,64) and sepsis-induced muscle atrophy in C2C12 myotubes(65). In patients with CIM, two transcriptomic analyses have reported differential expression of the NLRP3 gene(66) and functional enrichment of the Gene Ontology category "NLRP3 inflammasome complex"(67) in muscle biopsies from the tibialis anterior and vastus lateralis, respectively. In murine models of denervation and sepsis, NLRP3-associated muscle atrophy appears to be mediated by the upregulation of the E3 ubiquitin ligases MuRF1 and Atrogin-1, with NLRP3 gene deletion conferring a protective effect (68,69). The upregulation of these ligases is well documented in human CIM(12,40,42,66,70-73) and in various experimental models of this myopathy(74-82). Additionally, increased expression of other skeletal muscle E3 ligases, such as MUSA1(66,73), TRIM62(73), and TRIM32(66), has been described. This upregulation is associated with enhanced proteasome activity in muscle samples from critically ill patients with muscle atrophy. (42,71,83). Taken together, evidence

from murine models of denervation and sepsis indicates that the NLRP3 inflammasome contributes to muscle atrophy via upregulation of the UPS(68,69). Since these models replicate key features of CIM and increased NLRP3 gene expression has been reported in patients with CIM, it is plausible to propose that the NLRP3 inflammasome contributes to muscle atrophy in human CIM.

# 1.4.NLRP3 Inflammasome Activation in CIM: Priming and Oligomerization

Canonical activation of the NLRP3 inflammasome occurs in two steps. The first signal, known as "priming," is triggered by the detection of pathogen-associated molecular patterns (PAMPs) or damage-associated molecular patterns (DAMPs) via Toll-like receptors (TLRs), or through the activation of tumor necrosis factor-alpha (TNF- $\alpha$ ) and interleukin-1 $\beta$  (IL-1 $\beta$ ) receptors(57). This in turn activates the nuclear factor kappa B (NF- $\kappa$ B), which upregulates the transcription of NLRP3, pro-IL-1 $\beta$ , and pro-IL-18(57,84,85).

Given that the NLRP3 inflammasome can be activated by various inflammatory and pathogen-associated stimuli(85,86), and that sepsis and SIRS are common risk factors for CIM(4,25–27,29,32,87), the critical illness environment provides favorable conditions for priming. Supporting this notion, increased expression of TNF- $\alpha$ , TNFR, and IL-1 $\beta$  has been reported in the muscle tissue of patients with CIM(40,66,71,73,88), as well as in murine models of sepsis (89).

Moreover, overexpression of genes related to the NF-kB signaling pathway has been documented in skeletal muscle from patients with CIM(90) and in a murine ICU model(77), suggesting a potential pivotal role of this transcription factor in CIM pathogenesis. Therefore, it is reasonable to hypothesize that priming of the NLRP3 inflammasome may occur during the development of CIM.

Regarding the second activation signal, or the assembly of the NLRP3 inflammasome complex, this also occurs in response to PAMPs and DAMPs (57,84,85). Oligomerization of the NLRP3 protein leads to the cleavage of pro-caspase-1, generating active caspase-1(57,85). This enzyme subsequently processes pro-IL-1 $\beta$  and pro-IL-18 into their active forms. Caspase-1 also cleaves gasdermin D (GSDMD), and the N-terminal fragment (GSDMD-NT) oligomerizes to form pores in the plasma membrane, facilitating the secretion of IL-1 $\beta$  and IL-18 and initiating inflammatory responses, including pyroptotic cell death (57,84,85,91).

A broad array of intracellular conditions and mediators contribute to this second activation step(57,84,85). Among them, mitochondrial dysfunction and the production of reactive oxygen species (ROS) are considered major stimuli for NLRP3 inflammasome activation(92-94). Mitochondrial dysfunction is well documented in critical illness and during the early stages of CIM(38). This has been evidenced by: (a) disruption of mitochondrial ultrastructure (89,95–99); (b) dysregulation of mitochondrial biogenesis factors—such as TFAM(95,98-100), TFBM1, TFBM2(98–100), PGC1 $\alpha$ (42,88,95,96,98,100–103), PGC1 $\beta$ (100), PPAR $\gamma$ 2(82), PPRC1(102), NRF-1(95,98,100), and NRF-2(98,100,101); (c) increased mitophagy as indicated by elevated Bnip3 expression(40,70,72,76,98,104); (d) reduced ATP synthesis and oxidative phosphorylation(88,89,105,106); (e) alterations in levels, expression, and activity of mitochondrial respiratory complexes (79,80,95-97,99-101,103,106-108); (f) redox imbalance reflected by changes in superoxide dismutase levels and reductions in various antioxidant enzymes(51,95,99,100,103,104); and (g) increased oxidative stress, as shown by lipid peroxidation, protein carbonylation, and nitration(70,97,100,103,109). Taken together, these findings support the hypothesis that activation and assembly of the NLRP3 inflammasome may occur in human CIM. Additionally, the release of lysosomal contents such as cathepsin B also contributes to this second signal and NLRP3 inflammasome assembly (85,110). In CIM, increased expression and activity of cathepsin L(40,70,72) and cathepsin B(66,72), among others(66), have been reported, along with an increased presence of lysosomal vacuoles and vesicles(13,70). Therefore, mitochondrial dysfunction, oxidative stress, and elevated cathepsin activity—features described in CIM—may be mechanistically linked to the second activation signal of the NLRP3 inflammasome. However, this association has not yet been specifically studied in CIM.

# 1.5.Physical Therapy, Inflammation, and Potential Modulation of the NLRP3 Inflammasome in CIM

Mechanical silencing due to prolonged bed rest is a key risk factor in the development of CIM. Importantly, this factor is modifiable through early mobilization(4,25,27–29,31). However, further evidence is needed to support the notion that physical therapy(3,111), active mobilization, and rehabilitation in critically ill patients can improve muscle strength and functional status. These interventions may reduce the incidence of CIM and shorten hospital stays(3,4,25,112–116).

Physical therapy has demonstrated biological effects on the muscles of critically ill patients, as well as in experimental models of CIM. In a murine ICU model, physical therapy was shown to exert a protective effect against myosin loss, while increasing the expression of sarcomeric proteins and growth factors involved in muscle development (80). Kalamgi et al. reported that physical therapy increased levels of Akt, p-Akt, p-S6, as well as the expression of myogenin and MyoD(76), suggesting that mobilization promotes protein synthesis and muscle repair pathways in murine models of critical illness. In a randomized controlled trial, Hickmann et al. described a reduction in REDD1 expression(40), which may enhance mTOR signaling and protein synthesis(117). The same study reported decreased expression of Bnip3, Gabarapl1, and Lc3b, and increased p-ULK1<sup>Ser757</sup>, a condition that inhibits autophagy. Additionally, the authors observed reduced colocalization of p62 with Lamp-2A(40), suggesting a decrease in chaperone-mediated autophagy. In a murine ICU model, mechanical loading was found to induce PGC-1α4 (an exercise-induced isoform)(76), thereby promoting mitochondrial biogenesis. Based on current evidence, physical therapy and early mobilization in critically ill patients may exert effects on mitochondrial function and autophagy, potentially influencing NLRP3 inflammasome activation. However, this regulatory role has not yet been demonstrated in the skeletal muscle of critically ill patients with CIM. Regarding physical therapy and its relationship with systemic inflammation, several studies have described its modulatory effect on the inflammatory state across different health conditions (118–132). arious forms of exercise and physical therapy have been shown to reduce levels of IL- $1\beta(124,131,132)$  and TNF- $\alpha(124,128,130)$  in multiple pathologies. In elderly populations, exercise reduces levels of NLRP3 and caspase-1(133). Furthermore, physical therapy and exercise have been associated with reduced NLRP3 inflammasome activity in murine models of Parkinson's disease(134); post-stroke depressio(135); and chronic kidney diseaseassociated cachexia(136) Similarly, in a murine model of sciatic nerve injury, decreased levels of IL-1 $\beta$  and TNF- $\alpha$  were observed(137). However, the potential modulatory effect of physical therapy on the NLRP3 inflammasome and its role in the development of CIM has not yet been described. The pathogenesis of inflammation-associated muscle atrophy remains unclear (84). particularly in CIM. Therefore, understanding the molecular mechanisms underlying this condition is of great importance.

In summary: (1) Skeletal muscle from patients with CIM shows overexpression of the NLRP3 inflammasome gene and associated signaling components; (2) the NLRP3 inflammasome promotes muscle atrophy through upregulation of atrogenes in murine models of sepsis, denervation, and in C2C12 myotubes; (3) critically ill patients exhibit systemic inflammation, sepsis, and elevated levels of TNF- $\alpha$  and IL-1 $\beta$ —conditions that promote NLRP3 inflammasome priming; (4) CIM is characterized by mitochondrial dysfunction, oxidative stress, and increased cathepsin B, all of which favor the second activation signal of the NLRP3 inflammasome; (5) in various pathological contexts, physical therapy has been shown to reduce inflammation, IL-1 $\beta$ , TNF- $\alpha$ , and NLRP3 inflammasome levels, suggesting it may act as a protective factor against NLRP3-mediated muscle atrophy in CIM.

Based on these observations, the following research questions arise: In human CIM: (a) Is NLRP3 inflammasome activation associated with muscle atrophy via upregulation of atrogenes?; (b) Does physical therapy reduce NLRP3 inflammasome activation in the skeletal muscle of patients with CIM, thereby contributing to the attenuation of muscle atrophy?

Figure 1 provides a graphical summary of the proposed contribution of the NLRP3 inflammasome to muscle atrophy in CIM, and the potential protective effect of physical therapy.



Figure 1. Proposed contribution of the NLRP3 inflammasome to muscle atrophy in critical illness myopathy and the protective effect of physical therapy.

Based on the aforementioned background, the hypothesis of this research project is:

#### 2. Hypothesis

Physical therapy reduces NLRP3 inflammasome activity and mitigates muscle atrophy in critical illness myopathy.

# 3. General Objective

To investigate the association between the effects of physical therapy on NLRP3 inflammasome activation and muscle atrophy in critical illness myopathy.

# 4. Specific Objectives

- **4.1. SO1:** To evaluate the effect of physical therapy on NLRP3 inflammasome activation in vastus lateralis biopsies from patients with CIM, and to compare this activity with that of control patients.
- **4.2. SO2:** To assess the effect of physical therapy on muscle atrophy in vastus lateralis biopsies from CIM patients, and to relate these findings to NLRP3 inflammasome activation
- **4.3. SO3:** To determine the effect of physical therapy on the gene expression profile of signaling pathways involved in skeletal muscle atrophy in CIM patients.
- **4.4. SO4:** To analyze the association between gene expression and skeletal muscle biochemical parameters and the clinical diagnosis of CIM.

# 5. Experimental Design

SO1: To evaluate the effect of physical therapy on NLRP3 inflammasome activation in vastus lateralis biopsies from CIM patients, and to compare this activity with that of control patients.

**Rationale:** The NLRP3 inflammasome causes muscle atrophy in murine models of CIM (68,69). Prolonged bed rest, a major risk factor for CIM, is modifiable through physical therapy (4,25,27–29,31). This intervention has been shown to modulate inflammation(118–132) and the NLRP3 inflammasome(133), reduce levels of IL-1 $\beta$  and TNF- $\alpha$ (124,128), and influence mitochondrial function and autophagy(40), potentially leading to decreased inflammasome activation. However, this relationship has not been explored in human CIM. **Experimental approach:** Patients with CIM will be randomized to receive conventional or additional physical therapy. Non-CIM patients will serve as controls. From serum and vastus lateralis biopsies, the following will be assessed:

- 1. **NLRP3 inflammasome priming:** Protein levels of phospho-p65<sup>S536</sup> and total p65 will be measured via Western blot; mRNA levels of NLRP3, IL-1β, and IL-18 via RT-qPCR.
- 2. **NLRP3 inflammasome activity:** Cleaved IL-1β, cleaved caspase-1, and GSDMD-NT will be quantified by Western blot relative to their precursor forms. IL-1β and IL-18 levels in plasma will be measured by ELISA.
- 3. **Second-signal activation factors:** Oxidative stress markers (protein carbonylation and nitration) and cathepsin B levels will be evaluated by Western blot and RT-qPCR. In addition, mitochondrial ultrastructure and the presence and volume of lysosomal vacuoles will be analysed by transmission electron microscopy as a strategy to assess mitochondrial dysfunction and dysregulated autophagy.

**Expected outcomes:** Physical therapy is expected to reduce NLRP3 inflammasome activation in a frequency- and duration-dependent manner.

**Pitfalls:** If difficulties arise in measuring the proposed signaling pathway from muscle biopsy lysates, primary skeletal muscle cultures will be used to study inflammasome activity. Caspase-1 activity will also be assessed using a fluorometric kit (FAM-FLICA™, Bio-Rad).

SO2: To assess the effect of physical therapy on muscle atrophy in vastus lateralis biopsies from CIM patients, and to relate these findings to NLRP3 inflammasome activation.

**Rationale:** Muscle mass loss in CIM is partly attributed to atrogene overexpression(7). In murine models, NLRP3 contributes to atrophy through this mechanism (68,69). However, this association—and its modulation by physical therapy—has not yet been explored in humans. **Experimental approach:** The characteristics of CIM and muscle atrophy will be correlated with findings from SO1:

- Muscle atrophy: Muscle cryosections (10 μm) will be analyzed by indirect immunofluorescence using anti-laminin to delineate cell boundaries and quantify fiber diameter. mRNA levels of atrogenes—MuRF1, Atrogin-1, MUSA1, TRIM62, and TRIM32—will be measured by RT-qPCR.
- 2. **Molecular and histological features of CIM:** Myosin/actin ratio will be quantified by Western blot using biopsy homogenates. Sarcomeric organization will be evaluated in 10 µm cryosections using transmission electron microscopy.

**Expected outcomes:** Physical therapy is expected to reduce muscle atrophy in relation to intervention frequency and duration. These effects are expected to be associated with changes in NLRP3 inflammasome activation.

**Pitfalls:** If the proposed evaluations are not feasible, miRNA expression related to muscle atrophy will be assessed via nanopore sequencing. If immunofluorescence is not possible, myofiber cross-sectional area will be analyzed using H&E histology.

SO3: To determine the effect of physical therapy on the gene expression profile of signaling pathways involved in skeletal muscle atrophy in CIM patients. Rationale: Transcriptomics has advanced rapidly in critical care, enabling early diagnosis, precision medicine (138,139), and identification of key signaling pathways associated with gene expression changes (138,140). Such analyses have been applied in CIM patients (66,67,141),

and murine models(76,80,142). However, only one study has investigated the effect of physical therapy on transcriptomics in CIM, and it did not show significant effects, likely due to its sample size and unilateral intervention(66). More studies are needed to uncover the underlying mechanisms of CIM and the impact of early mobilization.

**Experimental approach:** Differential gene expression related to NLRP3 inflammasome and skeletal muscle atrophy pathways will be assessed via microarray. **Expected outcomes:** Greater differential expression of genes associated with muscle atrophy is expected in CIM patients. Physical therapy is expected to modulate this expression. **Pitfalls:** If technical or interpretative issues arise with the microarray, mRNA sequencing will be performed using nanopore technology.

# SO4: To analyze the association between gene expression and skeletal muscle biochemical parameters with the clinical diagnosis of CIM.

**Rationale:** Early diagnosis of CIM is crucial. Although tools like the SOFA score and muscle ultrasound have shown promise(39,40), more evidence is needed to validate their use(41). **Experimental approach:** Molecular biology findings and gene expression profiles will be associated with the clinical and ultrasound-based diagnosis of CIM, in conjunction with critical illness severity, to support early detection strategies.

**Expected outcomes:** A strong association is expected between early CIM diagnosis, clinical markers, and biochemical/histological findings.

#### 6. Patients and Methods

# 6.1.Study Design

This pilot study adopts a quantitative approach, with an analytical, experimental, prospective, and longitudinal design.

#### 6.2. Patients

# 6.2.1. CIM Patients (Group A, n = 16)

**Inclusión Criteria:** Critically ill patients with CIM will be selected based on the following inclusion criteria:

- 1. Medical diagnosis of sepsis upon ICU admission,
- 2. Receiving invasive mechanical ventilation with a projected requirement ≥7 days,
- 3. SOFA score ≥8 for three consecutive days within the first five days of ICU admission (22.41.42.81.141.144).

To screen for CIM in these patients, serial quadriceps ultrasound assessments will be conducted at three timepoints: within the first 24 hours of ICU admission, again within the first 72 hours, and finally 7 days after the second assessment. The ultrasound protocol is detailed in Annex 2. Changes in muscle thickness, cross-sectional area, pennation angle, and echogenicity will be evaluated. Patients meeting the following criteria within 7–10 days of ICU admission will be considered suspected CIM cases:  $\geq$ 20% reduction in muscle thickness,  $\geq$ 10% reduction in cross-sectional area,  $\geq$ 5% decrease in pennation angle,  $\geq$ 8% increase in echogenicity(37).

For patients who regain consciousness and are cooperative, muscle strength will be assessed using the Medical Research Council Sum Score (MRC-SS); a score ≤48 confirms muscle weakness(9,33,145).

Exclusion criteria: Patients will be excluded if they present with: neurocritical illness, prior malnutrition or cachexia, pre-existing neuromuscular disease, coagulopathy (severe liver disease or continuous dialysis), thrombocytopenia <20,000 platelets/μL, inability to walk independently prior to hospitalization or low pre-admission functional status (Clinical Frailty Scale ≥4), lower limb amputation, lower limb fractures, ongoing chemotherapy, pregnancy, BMI >35, uncontrolled epilepsy, allergy to ultrasound gel, prolonged corticosteroid therapy, expected ICU stay <7 days, imminent death, or legal guardian refusal to provide informed consent.

# **Group A Subgroups:**

- A.1: CIM patients receiving conventional physical therapy
- A.2: CIM patients receiving additional physical therapy (servo-assisted lower limb mobilization using Motomed Letto® at 30 rpm, 2 sessions/day, 60 minutes/session for 7 days).

Although no specific treatment exists for CIM(66), prior studies have evaluated the effect of prolonged physical therapy compared to standard care (40,66), allowing all patients access to this intervention regardless of standardization(40,147,148). Therapy dosage may be titrated by adjusting rpm intensity, under safety criteria defined by Hodgson's expert consensus(149) and continuous monitoring of hemodynamic and respiratory parameters.

# 6.2.2. Control Patients (Group B, n = 8)

Control patients will be recruited from those admitted for conditions unrelated to CIM and who are conscious and capable of providing informed consent.

**Exclusion criteria:** Same as for Group A, with the addition of: laboratory evidence of systemic inflammation (elevated C-reactive protein and/or leukocytosis) and refusal to consent.

#### 6.2.3. Patient Recruitment Sites

All Group A and B patients will be recruited from the Adult Critical Care Unit at the Hospital de Urgencia y Asistencia Pública (Ex Posta Central) and Clínica INDISA. Each participant will have a clinical file where all morbidity data will be recorded. Either the patient or their legal guardian will sign an informed consent form outlining all study procedures. All information will be treated with strict confidentiality.

# 6.3. Sample Size Validation

The sample size was calculated based on the increased gene expression of IL-1 $\beta$  observed in vastus lateralis muscle biopsies from critically ill patients with sepsis, reported as 15.36 times higher than that of healthy controls (with a standard deviation of 4.96), according to Hickmann et al.(40). This expression level is proposed as the effect size, or the variable to be reduced by physical therapy, under the assumption that IL-1 $\beta$  gene expression reflects NLRP3 inflammasome activation in skeletal muscle.

Assuming a statistical power of 99%, a type I error (alpha) of 5%, and an anticipated 40% mortality rate in critically ill patients (to account for potential loss)(150), the estimated sample size was 8 patients with CIM per physical therapy group. Based on the principle of equivalence, the control group will also include 8 patients. Sample size was calculated using R Studio with the following command: n.ttest(power = 0.99, alpha = 0.05, mean.diff = 15.36, sd1 = 4.96, design = "unpaired", variance = "unequal").

# 6.4. Sample Collection from Patients with CIM and Controls

# 6.4.1. Vastus Lateralis Muscle Biopsy

Two samples of the vastus lateralis muscle will be obtained from both CIM patients and controls: the first within the initial 3 days of ICU admission, and the second 7 days later. The muscle biopsy procedure is well-established in the literature (12,13,39,40,42,49,67,71–73,81–83,88,95,99,101,104–106,141,144,151). A percutaneous needle biopsy (TPNB) will be used, as it is a minimally invasive technique(152) that has demonstrated good yield in critically ill patients for gene expression, protein, and ultrastructural analyses(40). Under local anesthesia with 2% lidocaine, three to five samples of the vastus lateralis (VL) muscle will be collected using a disposable 12-gauge coaxial biopsy needle (BARD, MAGNUM®) to obtain approximately 90 mg of tissue. The first sample will be taken at a 90° angle and stored at -80°C for histological studies. The remaining samples will be cleared of blood with sterile gauze, snap-frozen in liquid nitrogen, and stored at -80°C for gene and protein expression analysis.

# 6.4.2. Blood Samples

Each CIM patient and control subject will donate 10 ml of peripheral blood on two occasions, collected in EDTA vacutainers (Becton Dickinson Ind Cir Ltda.) as anticoagulant. The sampling will be synchronized with the timing of muscle biopsy collection.

# 6.5. Evaluators

The methodology requires ultrasound assessment of the quadriceps muscle and the use of the MRC Sum Score and FSS-ICU scales by physical therapists from the ICU. Although these professionals have clinical experience with these evaluations and adequate inter-rater reliability has been reported in the literature(145,153–158), it is necessary to verify inter-evaluator concordance. A prior pilot study titled "Validation of Operators and Inter-Evaluator Variability in Diagnostic Strategies for ICU-Acquired Weakness" will be conducted in cooperative patients capable of providing consent. This study is under development and has received ethical approval from the Scientific Ethics Committee of Clínica INDISA (Protocol No. 176-25-24).

# 6.6. Histological and Biochemical Methods

# 6.6.1. Histology

Transmission electron microscopy (TEM) will be performed on ultrathin 10  $\mu$ m cryosections from muscle biopsy fragments. Sections will be fixed in 2.5% glutaraldehyde for 2 hours at room temperature, washed four times in 0.1 M sodium cacodylate buffer, dehydrated in graded acetone series, and embedded in Epon resin. Ultrathin sections will be contrasted sequentially with 2% osmium tetroxide in 0.1 M sodium cacodylate buffer and 1% uranyl acetate in the same buffer, then examined via TEM.

#### 6.6.2. Immunofluorescence

10 µm cryosections will be washed with TBS-T (Tris-buffered saline with 0.1% Tween20®), fixed with 100% cold acetone for 30 minutes at -20°C, then blocked with 3% BSA in TBS-T for 2 hours. Permeabilization will be performed using 0.1% Triton X-100 in 3% BSA for 30 minutes. Primary antibody against laminin (1:30, L9393, Sigma-Aldrich) will be incubated overnight at 4°C, followed by secondary antibody Alexa Fluor 488 Goat anti-Rabbit (1:500, Life Technologies) for 2 hours at room temperature in the dark. Slides will be mounted with ProLong containing DAPI (Life Technologies), stored at 4°C, and imaged by confocal microscopy. Muscle fiber diameter will be measured using ImageJ software and compared against control values to determine muscle atrophy.

# 6.6.3. Western Blot

30 mg of muscle biopsy samples will be lysed using an automated homogenizer (D1000, Biolab, Madrid, Spain) in a lysis buffer containing: 1X T-PER (#78510, ThermoFisher, Massachusetts, USA), 1 mM EGTA (Winkler, Santiago, Chile), 1 mM EDTA (Winkler, Santiago, Chile), 2 mM BAPTA (#A4926, Sigma Aldrich, Missouri, USA), 10 mM NaVO<sub>4</sub> (#S6508, Sigma Aldrich, Missouri, USA), 10 mM Na<sub>2</sub>P<sub>2</sub>O<sub>7</sub> (Winkler, Santiago, Chile), 1X protease inhibitor (#04693124001, Roche, Mannheim, Germany) and 1X phosphatase inhibitor (#04906845001, Roche, Mannheim, Germany). Samples will then be centrifuged at 4°C for 14 minutes at 12,000 rpm. The supernatant will be analyzed by SDS-PAGE (8% or 10%, depending on the target protein). Wet electrotransfer will be performed onto polyvinylidene fluoride (PVDF) membranes, which will be blocked with 5% semi-skimmed milk (SVELTY®) in TRIS-buffered saline with 0.1% Tween 20 (TBS-T), followed by TBS-T washes. Membranes will be incubated with the primary antibody for 16 hours at 4°C. Subsequently, incubation with the appropriate HRP-conjugated secondary antibody will be carried out—either anti-rabbit (1:10,000, 7074, Cell Signaling) or anti-mouse (1:10,000, 516102, Santa Cruz Biotechnology). Membranes will be developed using enhanced chemiluminescence (ECL) reagent (sc-2048, Santa Cruz Biotechnology), and images will be acquired with the LI-COR C-Digit imaging system and Image Studio software (Lincoln, Nebraska, USA). Individual protein levels and protein-toprotein ratios will be compared with those obtained from control patients without neuromusculoskeletal disease.

#### 6.6.3.1. Myosin/Actin Ratio

Membranes will be incubated with two antibodies: anti-myosin antibody diluted 1:1000 (F59: sc-32732, Santa Cruz Biotechnology), and anti-actin antibody diluted 1:1000 (HUC1-1: sc-53141, Santa Cruz Biotechnology). The myosin/actin ratio will then be calculated. A ratio below 1.5 is considered conclusive for myopathy (6,12,13,90).

# 6.6.3.2. Priming of the NLRP3 Inflammasome

To assess the phosphorylation levels of p65 (a component of the NF-κB complex), membranes will be incubated with two antibodies: anti-p65S536 antibody diluted 1:1000 (sc-101752, Santa Cruz Biotechnology) and total anti-p65 antibody diluted 1:1000 (sc-8008, Santa Cruz Biotechnology).

# 6.6.3.3. Activation of the NLRP3 Inflammasome

To evaluate the activation of the NLRP3 inflammasome, the ratios of cleaved caspase-1/procaspase-1, cleaved IL-1 $\beta$ /pro-IL-1 $\beta$ , and GSDMD-N/GSDMD will be determined.

# 6.6.3.3.1. Cleaved Caspase-1/Pro-Caspase-1 Ratio

Membranes will be incubated with two antibodies: anti-cleaved caspase-1 antibody diluted 1:1000 (4199, Cell Signaling) and anti-caspase-1 antibody diluted 1:1000 (3866, Cell Signaling).

# 6.6.3.3.2. Cleaved IL-1β/Pro-IL-1β Ratio

Membranes will be incubated with two antibodies: anti-cleaved IL-1β antibody diluted 1:1000 (83186, Cell Signaling) and total anti-IL-1β antibody diluted 1:1000 (12703, Cell Signaling).

#### 6.6.3.3.3. GSDMD-N/GSDMD Ratio

Membranes will be incubated with two antibodies: anti-GSDMD-N antibody diluted 1:1000 (ab215203, Abcam) and anti-GSDMD antibody diluted 1:400 ((H-11): sc-393581, Santa Cruz Biotechnology).

# 6.6.3.4. Secondary Activation of the NLRP3 Inflammasome

To assess conditions that favor the secondary activation of the NLRP3 inflammasome, oxidative stress and increased cathepsin B due to dysregulated autophagy will be evaluated. Oxidative stress will be assessed by measuring protein carbonylation and nitration. Protein carbonylation will be detected using the OxyBlot™ Protein Oxidation Detection Kit (EMD Millipore), according to the manufacturer's instructions. Protein nitration will be assessed using anti-nitrotyrosine antibody diluted 1:2000 ((39B6): sc-32757, Santa Cruz Biotechnology). Cathepsin B levels will be quantified using anti-cathepsin B antibody diluted 1:1000 (H-5: sc-365558, Santa Cruz Biotechnology). GAPDH will be used as a loading control, detected with anti-GAPDH antibody diluted 1:2000 ((0411): sc-47724, Santa Cruz Biotechnology).

# 6.6.4. RT-qPCR

A total of 20 mg of muscle biopsy tissue will be lysed using an automatic homogenizer (D1000, Biolab, Madrid, Spain) in 1 mL of TRIzol reagent (Invitrogen). The lysate will be incubated at room temperature for 5 minutes to ensure complete dissociation of nucleoprotein complexes. Then, 200  $\mu L$  of chloroform per mL of TRIzol will be added to the homogenate tubes and vigorously shaken for 30 seconds. After 2–3 minutes of incubation, the samples will be centrifuged at 12,000 g for 15 minutes at 4°C. The aqueous phase will be transferred to a new microcentrifuge tube. To precipitate RNA, 200  $\mu L$  of isopropanol per 1 mL of TRIzol used will be added and incubated for 2 hours at -20°C. The samples will then be centrifuged at 12,000 g for 10 minutes at 4°C, and the supernatant will be discarded. For RNA washing, the pellet will be suspended in 1 mL of 75% ethanol at -20°C (same volume of TRIzol used for lysis), briefly vortexed, and centrifuged at 7500 g for 5 minutes at 4°C. After discarding the supernatant, the RNA pellet will be air-dried for 5–10 minutes. To solubilize the RNA, the pellet will be resuspended in 20–30  $\mu L$  of RNase-free water and incubated on a heat block at 55–60°C for 10–15 minutes. RNA concentration will be measured using the MaestroNano spectrophotometer.

Reverse transcription will be performed using the iScript cDNA Synthesis Kit (Bio-Rad). Reactions will be carried out in a final volume of 10  $\mu$ L containing 1  $\mu$ g of RNA, 0.1  $\mu$ L of each primer (100 nM final), and 5  $\mu$ L of cDNA. Thermal cycling will follow this protocol: 3 minutes at 95°C, followed by 40 cycles of 30 seconds at 95°C, 30 seconds at 60°C, and 30 seconds at 72°C. SYBR® Green (Applied Biosystems) will be used as the fluorescent probe. All samples will be run in duplicate.  $\beta$ 2-microglobulin ( $\beta$ 2M) will be used as the reference gene, as it has shown stable expression levels regardless of the exercise modality (159).

#### 6.6.4.1. Priming of the NLRP3 Inflammasome

To assess the priming of the NLRP3 inflammasome, RT-qPCR will be performed to quantify mRNA levels of NLRP3, IL-1 $\beta$ , and IL-18.

# 6.6.4.2. Secondary Activation of the NLRP3 Inflammasome

To evaluate dysregulated autophagy favoring the secondary activation of the NLRP3 inflammasome, RT-qPCR will be used to assess Cathepsin B mRNA expression.

# 6.6.4.3. Atrogenes

To evaluate the ubiquitin-proteasome system, RT-qPCR will be performed to quantify mRNA levels of the ubiquitin ligases: MurF1, Atrogin-1, MUSA1, TRIM62, and TRIM32.

#### Primer List:

| = | | |
|---|---|---|
| Gene | Forward Primer | Reverse Primer |
| NLRP3 | 5'-GAGGAAAAGGAAGGCCGACA-3' | 5'-CCCGGCAAAAACTGGAAGTG-3' |
| IL-1β | 5'AGCAACAAGTGGTGTTCTCCATGT-3' | 5'-AGCTGTAGAGTGGGCTTATCATCTT-3' |
| IL-18 | 5'-AGCCTAGAGGTATGGCTGTAAC-3' | 5'-AAAGGTCTCTCTCTTTTTCACAAGC-3' |
| Catepsina B | 5'-GCGCTGGGTGGATCTAGGA-3' | 5'-GTTGACCAGCTCATCCGACA-3' |
| MurF1 | 5'-AAACAGGAGTGCTCCAGTCGG-3' | 5'-CGCCACCAGCATGGAGATACA-3' |
| Atrogina-1 | 5'-CGACCTCAGCAGTTACTGCAA-3' | 5'-TTTGCTATCAGCTCCAACAG-3' |
| MUSA1 | 5'-GTGATCATGCCAATCCACAG-3' | 5'-CATGAATGTCACCATGCACA-3' |
| TRIM62 | 5'-AAGTCCCTGTTCCAGGACATC-3' | 5'-GCAGTCGTCCGACAGGAT-3' |
| TRIM32 | 5'-CCCCATAGGGGATGAGAAAT-3' | 5'-GTCCTATTTGGGCAGTGCAT-3' |
| Fbxo21/SMART | 5'-CACGTTCCTTGTAATGGCTTCA-3' | 5'-ACGACTCATAGTCATCTGGCTG)-3' |
| β2M (Housekeeping) | 5'-ATGAGTATGCCTGCCGTGTGA-3' | 5'GGCATCTTCAAACCTCCATG-3' |

# 6.6.5. ELISA

EDTA vacutainer tubes will be centrifuged for 10 minutes at 4°C and 4000 rpm. Plasma and serum will be aliquoted into microcentrifuge tubes with 500  $\mu$ L per sample. Measurements will be performed according to the manufacturer's instructions using the following kits: IL-1 $\beta$ : Human IL-1 $\beta$  ELISA Kit (Invitrogen), IL-18: Human IL-18 ELISA Kit (Invitrogen).

# 6.6.6. Microarray.

Total mRNA will be extracted from samples of control and CIM (Critical Illness Myopathy) patients. Using reverse transcriptase (RT), complementary DNA (cDNA) libraries will be synthesized from the extracted RNA. These cDNA libraries will be labeled with fluorescent probes incorporated during synthesis. The labeled cDNA samples will then be hybridized to a commercial microarray chip containing oligonucleotides with complementary sequences. This hybridization process results in a stable DNA double helix. After hybridization, the chip will be washed several times to remove any unbound cDNA. The chip will then be scanned using a laser to excite the fluorescent tags. The fluorescence signal from each spot will be captured and analyzed with specialized software that generates a colorimetric image of the microarray. Expression profiles will be obtained using Illumina HT-12 v4 microarrays (one microarray per sample).

# 6.6.6.1. Microarray Data Analysis

Raw expression data will be processed using the R software environment and the "Bioconductor" package. The data will undergo background correction, quantile normalization, and log2 transformation using the neqc function from the *limma* package. Probes classified as "No match" or "Bad" will be removed using the *illuminaHumanv4* annotation package.

# 6.6.6.2. Differential Gene Expression

Robust differential expression analysis of all probes will be performed using the *limma* package in R, adjusted for each patient's sociodemographic and clinical variables. Sample correlation will be assessed using the duplicateCorrelation function. The decideTests function with the "global" adjustment will be used to estimate the false discovery rate (FDR), using a significance threshold of FDR < 0.05 and a minimum expression change of 1.5-fold compared to controls.

# 6.6.6.3. Gene Ontology (GO)

Functional enrichment analysis in Gene Ontology will be performed using the "gProfiler" tool in R. The statistical threshold for GO enrichment will be an FDR-adjusted p-value < 0.05, with a minimum of 10 detected genes. The enrichment list will include all genes represented in the Illumina Human HT-12 v4 array with a p-value < 0.05 in at least three samples.

# 6.7.Demographic Variables, Severity of Critical Illness, Clinical Assessment of Muscle Strength, and Functionality

The sociodemographic and clinical variables that will be recorded throughout the study include: biological sex, age, body mass index (BMI), degree of hypoxemia, comorbidities, route of nutrition, nitrogen balance, serum albumin, lactatemia, duration of mechanical ventilation, length of ICU stay, and total hospitalization. The severity of critical illness will be assessed using the SOFA (Sequential Organ Failure Assessment) score. The use and dosage of the following medications will also be recorded: norepinephrine, milrinone, dobutamine, propofol,

ketamine, midazolam, dexmedetomidine, neuromuscular blocking agents, corticosteroids, and aminoglycosides.

Regarding physical therapy and functionality, the Clinical Frailty Scale(160) will be used to determine the functional status prior to ICU admission. In cooperative patients (those who respond to at least 3 out of 5 commands in the S5Q scale—five standardized ICU questions), analytical muscle strength will be assessed using the Medical Research Council Sum Score (MRC-SS)(9,33,145). A score of ≤48 points confirm the presence of muscular weakness, which must be corroborated by ultrasound and SOFA scale findings. This scale also allows for the classification of severe muscle weakness when the score is below 36 points(33,34,41). Functional status will be assessed using the Functional Status Score for the ICU (FSS-ICU)(46,158,161). Data collection will include the time elapsed until the first physical therapy session, the number of sessions, the modality of intervention, and its temporal distribution.

# 6.8. Statistical Analysis

Primary quantification results will be expressed as gene or protein expression levels relative to control patients. These will be reported using central tendency and dispersion measures, and normality will be assessed using the Shapiro–Wilk test.

For comparisons between independent groups, Student's t-test or the Wilcoxon rank-sum test will be applied, depending on the distribution of the data. To assess differences before and after the early physical therapy intervention, paired Student's t-tests or Wilcoxon signed-rank tests will be used.

Correlation between the outcome variables of Objective 1 (SO1) and Objective 2 (SO2) will be analyzed using Pearson or Spearman correlation coefficients, depending on variable distribution.

For differential gene expression analysis, quantification will be relative to control patients, and significance will be assessed with a false discovery rate (FDR) threshold of <0.05.

Associations between variables will be analyzed based on their nature. Multiple linear regression will be applied to quantitative variables. For associations between cellular and molecular biology findings and dichotomous variables (e.g., presence of muscle weakness), logistic regression will be used. For associations with ordinal variables, such as functional scales (e.g., FSS-ICU), Poisson regression will be applied. All statistical analyses and graph generation will be conducted using R Studio and Stata software.

# 7. Ethical Considerations

# 7.1.Social Utility

Critical illness myopathy (CIM) is a common cause of ICU-acquired weakness (ICUAW)(1). This condition is characterized by muscle atrophy and impaired contractility, both of which contribute to increased mortality(14–18), prolonged hospital stays (9,10,25,28), (extended durations of mechanical ventilation(19,20), elevated healthcare costs(9,10,29,31,44), and long-term physical disability(19,20). CIM may progress to post-intensive care syndrome (PICS), potentially resulting in persistent disability(4,28). A Chilean study reported that 40% of critically ill patients experience some degree of disability after hospital discharge(46). Therefore, understanding the etiology of CIM is essential for designing both pharmacological and non-pharmacological therapeutic strategies.

Several risk factors have been identified in the development of CIM(4.25), with prolonged immobility highlighted as a modifiable factor through physical therapy (4,25,27-29,31). This underscores the importance of evaluating the effects of physical therapy and supports the biomedical justification for dedicated clinical staff to manage and implement rehabilitation in critically ill patients. Since muscle protein degradation and electrophysiological abnormalities emerge within the first 10 days of ICU admission(39,40), early and timely rehabilitation is crucial. Early detection strategies for CIM are necessary. Internationally, research groups have implemented methods combining the Sequential Organ Failure Assessment (SOFA) score with ultrasound assessment to detect CIM in non-cooperative patients(22-24,41,42). While this method has proven effective in specialized research groups, it remains to be broadly adopted in Chile. Implementing this evaluation locally could facilitate early CIM detection and allow for better allocation of physical therapy resources, minimizing mechanical silencing — a modifiable risk factor. Currently, critical care units in Chile do not have full coverage for rehabilitation needs(162). Thus, biomedical research on CIM could benefit the general population by informing public policies that expand access to physical therapy and rehabilitation in intensive care units.

# 7.2. Protection of Vulnerable Groups

This study focuses on critically ill patients during the first days of admission to the intensive care unit (ICU), a population considered vulnerable due to the lack of consciousness resulting from sedoanalgesia. However, since the study specifically targets the development of critical illness myopathy (CIM), it can only be conducted in this population. The initial hospitalization period is when the risk factors associated with CIM development manifest (22,26,87,163). In accordance with Article 28 of Chilean Law No. 20.584, this study will include adult patients who "are physically or mentally incapable of expressing consent." It is important to note that "this physical or mental condition that prevents providing informed consent or expressing preference is a necessary characteristic of the target research population."

As such, the study protocol will be submitted for review by a scientific ethics committee. If approved, it will subsequently be submitted for evaluation to the Regional Health Authority (SEREMI). Once approved by these institutions, legal guardians will be approached to provide informed consent for the inclusion of patients in the research protocol. Furthermore, as stipulated by Article 28 of Law No. 20.584, once the patients have recovered from sedation, are cooperative, and demonstrate no delirium or physical incapacity, "consent or expression of preference will be sought from the individuals who have regained the physical or mental capacity to provide such consent or to express their preferences."

This research does not introduce any form of bias related to sex, race, or age among participants.

#### 7.3. Randomization

Patients at risk of developing CIM (Group A) who meet the inclusion criteria and do not fulfill any exclusion criteria will be randomly assigned to receive either conventional physical therapy or an enhanced physical therapy protocol using a servo-assisted lower limb cycling device (Motomed Letto®). This strategy has been employed in previous studies to assess the effects of physical therapy by comparing extended interventions with conventional protocols(40,66,146–148,164). This design ensures that all patients have access to early

physical therapy and rehabilitation, thereby avoiding comparison with a non-intervention group(40,147).

Randomization will be independent of ethnicity. However, in order to ensure homogeneity across intervention groups, stratification will be performed based on two factors: age and sex. Stratified randomization will be implemented, and allocation concealment will be applied only at the assignment stage. Due to the nature of the intervention—physical therapy—it will not be possible to blind either participants or investigators to the treatment received; thus, the study is classified as open-label.

Randomization will be conducted using R Studio software and the "randomizr" package. Stratification by age and sex will be performed using the "split" function.

#### 7.4.Adverse Events

This study involves performing a muscle puncture to obtain tissue samples from the vastus lateralis. This procedure is well established in the study of CIM (12,13,39,40,42,49,67,71–73,81–83,88,95,99,101,104–106,141,144,151). Although the most commonly used techniques for human muscle biopsy are the percutaneous needle biopsy (Bergström method)(49,67,70–72,82,83,99,101,106,151), conchotome(13,39,66), and Henckel-Tilley forceps(95,105), a more recently described method—tiny percutaneous needle biopsy (TPNB)—has shown advantages. This technique is less traumatic for patients(152) and has already been applied in CIM studies, providing adequate yield for gene expression, protein analysis, and ultrastructural studies without reports of adverse events(40).

The biopsy will be performed under local cutaneous anesthesia (2% lidocaine hydrochloride) with prior disinfection using topical chlorhexidine, employing a sterile technique and a coaxial disposable biopsy needle (BARD, MAGNUM®, C.R. Bard Inc., Covington, GA). To minimize the occurrence of adverse events, biopsies will be performed by intensivist physicians using ultrasound guidance, allowing image-assisted needle placement(165). In parallel, the clinical nurse of the intensive care unit, will supervise and provide nursing care for the biopsy sites.

As previously mentioned, patients at risk of CIM will be randomized to receive either conventional physical therapy or more frequent and prolonged sessions using a servo-assisted lower-limb cycling device (Motomed Letto®). Recent studies have demonstrated the safety of this type of intervention during physiotherapy in intensive care settings(147).

Ultrasound evaluation is routine in intensive care units(166). However, some cases of contact dermatitis due to ultrasound gel have been reported (167–172). Therefore, the skin of the area assessed by ultrasound will be monitored after each session. Additionally, the exclusion criteria in this protocol are designed to minimize the likelihood of adverse events.

#### 7.5.Benefit Assessment

Percutaneous muscle biopsy is recognized as an essential technique for advancing knowledge in muscle physiology and for the diagnosis of musculoskeletal disorders (165,173,174). Although general concerns exist regarding potential adverse events associated with this procedure, the incidence of complications is low and typically of minimal clinical relevance. The most commonly reported complications include pain, erythema, ecchymosis, edema, and bleeding (173). This study entails the inherent risks associated with muscle puncture; however, these are generally mild and self-limiting (173). The likelihood of significant complications is further reduced through the application of strict exclusion criteria.

In the event of a complication arising from the muscle biopsy procedure, medical professional liability insurance will be available to cover any associated harm. It is important to note that participants will not receive any direct clinical benefit from undergoing the biopsy procedure. This will be explicitly explained during the informed consent process to the legal guardians of the patients, and subsequently to the patients themselves, once they regain the cognitive capacity necessary to either continue with or withdraw from the study.

Physical therapy within the ICU is a standard intervention in critically ill patients and will be conducted in accordance with established safety criteria described in the literature (149). Additionally, an enhanced physical therapy regimen will be applied using servo-assisted cycling devices (147,148). Importantly, all enrolled patients will receive some form of physical therapy—either conventional or enhanced—thus ensuring that no participant is deprived of therapeutic benefit.

# 7.6. Protection of Privacy

All collected data will be securely stored under the custody of the principal investigator. Participant information will be recorded using the REDCap (Research Electronic Data Capture) platform. The presentation of study results will always preserve participant anonymity; no personal identifiers or sensitive data will be disclosed to third parties. Muscle biopsy samples will be processed at the Muscle Metabolism Laboratory, where they will remain under the custodianship of Dr. Paola Llanos Vidal.

# 7.7. Ethical Monitoring of the Project

Any issues that arise during the implementation of the study or any amendments to the protocol will be reported to the ethics committee. In accordance with Article 10 of Law 20.120, "Any serious adverse event occurring during the course of the research must be reported by the investigator to the Committee and to the Director of the institution where the research is being conducted."

# 7.8. Feasibility

This study is supported by the clinical teams of the Adult Intensive Care Units at the Hospital de Urgencia y Asistencia Pública (Ex Posta Central) and Clínica INDISA, which will serve as the recruitment centers from 2025 through the end of 2026.

The research project is led by Dr. Lilian Jara Sosa, Dr. Paola Llanos Vidal, and Dr. Denisse Valladares Ide. Dr. Lilian Jara Sosa is a geneticist with extensive experience in the field, including research on the genetic profile of myopathies in the Chilean population. Under her guidance, transcriptomic analyses and differential gene expression studies will be conducted using advanced sequencing and bioinformatics technologies.

Dr. Paola Llanos is a specialist in the activation pathway of the NLRP3 inflammasome in skeletal muscle in preclinical models of insulin resistance induced by obesity. She leads investigations focused on low-grade inflammation in skeletal muscle, employing biochemical, cellular, fluorescence and confocal microscopy techniques, as well as muscle fiber cultures.

Dr. Denisse Valladares Ide has extensive expertise in studying the molecular mechanisms underlying sarcopenia using human muscle biopsy samples. She is an active researcher on the modulatory role of physical activity on sarcopenia in elderly populations.

Experiments related to the quantification of markers of NLRP3 inflammasome "priming" and assembly, as well as transcriptomic analyses, will be carried out with funding from Fondecyt Regular Grant No. 1231103 awarded to Dr. Paola Llanos Vidal and Fondecyt Regular Grant No. 1241959 awarded to Dr. Denisse Valladares. The acquisition of the biopsy device and disposable 12-Gauge coaxial biopsy needles (BARD, MAGNUM®) will be financed through the operating expenses of the National Doctoral Scholarship ANID No. 21231808.

Additionally, the project has the formal approval of medical leadership and rehabilitation coordinators of the Adult Intensive Care Units at the Hospital de Urgencia y Asistencia Pública and Clínica INDISA.

The project also includes the participation of Dr. Margot Navarrete, physician, general surgeon and intensive care medicine resident, and Dr. Valentín López, physician and internal medicine specialist, who will be responsible for performing the muscle biopsies.

Clinical nurse Valentina Burgos will assist with the monitoring of the muscle biopsy puncture site and associated nursing care.

The complementary expertise of the thesis advisors, along with a multidisciplinary team, will allow the project to be developed with a translational (bench-to-bedside) approach.

# 8. Discussion

Why is it important to study Critical Illness Myopathy? CIM is a common condition among critically ill patients(17,31,43), associated with increased mortality (9,11,25,28,29,31), prolonged hospital stay(9,10,25,28), elevated healthcare costs, and reduced physical function and long-term quality of life(9,10,29,31,44). It may also lead to Post-Intensive Care Syndrome (PICS), characterized by persistent cognitive, mental, and physical dysfunction(4,28).

In this study, an increase in NLRP3 inflammasome activation is expected in critically ill patients, potentially contributing to muscle atrophy. NLRP3 inflammasome activation has been linked to the upregulation of muscle atrophy-related genes in established murine models of the disease(68,69). However, this relationship has not yet been described in human CIM. We hypothesize an association between changes in inflammasome activation and muscle atrophy in patients with CIM. This connection would be highly relevant, as muscle atrophy and impaired contractility are key features driving poor outcomes in these patients(14–20). While associations do not necessarily imply causation(3), the findings of this study, derived from ex vivo samples, may support a link between the proposed mechanism and CIM pathogenesis. This could lead to the identification of novel pharmacological and non-pharmacological therapeutic targets, including physical therapy.

Mechanical silencing due to prolonged bed rest is a major modifiable risk factor for the development of CIM(4,25,27–29,31). Physical therapy is a non-pharmacological intervention that could regulate the proposed mechanism of atrophy. This intervention has shown beneficial effects in both CIM patients and experimental models, particularly in improving mitochondrial function(40,76) and autophagy processes(40). Additionally, various modalities of exercise and physical therapy have been shown to reduce IL-1 $\beta$  and TNF- $\alpha$  levels in different pathological conditions(124,126,128,130–132,137). Therefore, physical therapy in critically ill patients could modulate NLRP3 inflammasome activation(57,84,85,91), and the associated muscle atrophy. However, to date, research groups studying CIM pathophysiology have not yet addressed the potential protective effects of physical therapy on this pathway.

As an additional methodological approach to evaluate the mechanisms involved in CIM development and the effects of physical therapy, a genetic screening strategy is proposed. Transcriptomic analyses have previously been performed in both CIM patients (66,67,82) and in murine models of this condition (76,80,142). Nevertheless, only one study has analyzed the impact of physical therapy in patients with CIM, reporting no significant changes in the skeletal muscle gene expression profile (66). It should be noted that this study included only 7 patients and compared one limb with the contralateral immobilized limb (66). In contrast, the present study proposes to assess the effects of conventional physical therapy versus additional physical therapy, as previously described in the literature (40,147). Given the scarcity of such studies and the rationale outlined in this project, there is a clear need to expand knowledge regarding the effects of early mobilization and the underlying mechanisms of CIM.

# 9. References

- 1. Z'Graggen WJ, Tankisi H. Critical Illness Myopathy. Journal of Clinical Neurophysiology. 2020 May;37(3):200–4.
- 2. De Jonghe B. Paresis Acquired in the Intensive Care Unit. A Prospective Multicenter Study. JAMA. 2002 Dec 11;288(22):2859.
- 3. Vanhorebeek I, Latronico N, Van den Berghe G. ICU-acquired weakness. Intensive Care Med. 2020 Apr 19;46(4):637–53.
- 4. Chen J, Huang M. Intensive care unit-acquired weakness: Recent insights. Journal of Intensive Medicine. 2024 Jan;4(1):73–80.
- 5. Kress JP, Hall JB. ICU-Acquired Weakness and Recovery from Critical Illness. New England Journal of Medicine. 2014 Apr 24;370(17):1626–35.
- 6. Schefold JC, Wollersheim T, Grunow JJ, Luedi MM, Z'Graggen WJ, Weber-Carstens S. Muscular weakness and muscle wasting in the critically ill. J Cachexia Sarcopenia Muscle. 2020 Dec 7;11(6):1399–412.
- 7. Wang W, Xu C, Ma X, Zhang X, Xie P. Intensive Care Unit-Acquired Weakness: A Review of Recent Progress With a Look Toward the Future. Front Med (Lausanne). 2020 Nov 23;7.
- 8. Barreiro E. Models of disuse muscle atrophy: therapeutic implications in critically ill patients. Ann Transl Med. 2018 Jan;6(2):29–29.
- 9. Fan E, Cheek F, Chlan L, Gosselink R, Hart N, Herridge MS, et al. An Official American Thoracic Society Clinical Practice Guideline: The Diagnosis of Intensive Care Unit–acquired Weakness in Adults. Am J Respir Crit Care Med. 2014 Dec 15;190(12):1437–46.
- Stevens RD, Marshall SA, Cornblath DR, Hoke A, Needham DM, de Jonghe B, et al. A framework for diagnosing and classifying intensive care unit-acquired weakness. Crit Care Med. 2009 Oct;37:S299–308.
- 11. Wilcox SR. Corticosteroids and neuromuscular blockers in development of critical illness neuromuscular abnormalities: A historical review. J Crit Care. 2017 Feb;37:149–55.
- 12. Derde S, Hermans G, Derese I, Güiza F, Hedström Y, Wouters PJ, et al. Muscle atrophy and preferential loss of myosin in prolonged critically ill patients\*. Crit Care Med. 2012 Jan;40(1):79–89.
- 13. Stibler H, Edström L, Ahlbeck K, Remahl S, Ansved T. Electrophoretic determination of the myosin/actin ratio in the diagnosis of critical illness myopathy. Intensive Care Med. 2003 Sep 1;29(9):1515–27.
- 14. Zhang XM, Chen D, Xie XH, Zhang JE, Zeng Y, Cheng AS. Sarcopenia as a predictor of mortality among the critically ill in an intensive care unit: a systematic review and meta-analysis. BMC Geriatr. 2021 Dec 2;21(1):339.
- 15. Yanagi N, Koike T, Kamiya K, Hamazaki N, Nozaki K, Ichikawa T, et al. Assessment of Sarcopenia in the Intensive Care Unit and 1-Year Mortality in Survivors of Critical Illness. Nutrients. 2021 Aug 8;13(8):2726.
- 16. Giani M, Rezoagli E, Grassi A, Porta M, Riva L, Famularo S, et al. Low skeletal muscle index and myosteatosis as predictors of mortality in critically ill surgical patients. Nutrition. 2022 Sep;101:111687.
- 17. Hrdy O, Vrbica K, Kovar M, Korbicka T, Stepanova R, Gal R. Incidence of muscle wasting in the critically ill: a prospective observational cohort study. Sci Rep. 2023 Jan 13;13(1):742.
- 18. Mayer KP, Thompson Bastin ML, Montgomery-Yates AA, Pastva AM, Dupont-Versteegden EE, Parry SM, et al. Acute skeletal muscle wasting and dysfunction predict physical disability at hospital discharge in patients with critical illness. Crit Care. 2020 Dec 4;24(1):637.
- 19. Rodriguez B, Larsson L, Z'Graggen WJ. Critical Illness Myopathy: Diagnostic Approach and Resulting Therapeutic Implications. Curr Treat Options Neurol. 2022 Apr 28;24(4):173–82.
- 20. Vongchaiudomchoke W, Sathitkarnmanee B, Thanakiattiwibun C, Jarungjitaree S, Chaiwat O. The association between sarcopenia and functional outcomes after

- hospital discharge among critically ill surgical patients. Asian J Surg. 2022 Jul:45(7):1408–13.
- 21. Friedrich O, Diermeier S, Larsson L. Weak by the machines: muscle motor protein dysfunction a side effect of intensive care unit treatment. Acta Physiologica. 2018 Jan;222(1):e12885.
- 22. Weber-Carstens S, Deja M, Koch S, Spranger J, Bubser F, Wernecke KD, et al. Risk factors in critical illness myopathy during the early course of critical illness: a prospective observational study. Crit Care. 2010;14(3):R119.
- 23. Vijayan D, Thomas SM, Rajagopal K. Association of SOFA Score with Severity of Muscle Wasting in Critically III Patients: A Prospective Observational Study. Indian Journal of Critical Care Medicine. 2023 Sep 30;27(10):743–7.
- 24. Nanas S, Kritikos K, Angelopoulos E, Siafaka A, Tsikriki S, Poriazi M, et al. Predisposing factors for critical illness polyneuromyopathy in a multidisciplinary intensive care unit. Acta Neurol Scand. 2008 Sep;118(3):175–81.
- 25. Tortuyaux R, Davion JB, Jourdain M. Intensive care unit-acquired weakness: Questions the clinician should ask. Rev Neurol (Paris). 2022 Jan;178(1–2):84–92.
- 26. Yang Z, Wang X, Wang F, Peng Z, Fan Y. A systematic review and meta-analysis of risk factors for intensive care unit acquired weakness. Medicine. 2022 Oct 28;101(43):e31405.
- 27. Schefold JC, Bierbrauer J, Weber-Carstens S. Intensive care unit—acquired weakness (ICUAW) and muscle wasting in critically ill patients with severe sepsis and septic shock. J Cachexia Sarcopenia Muscle. 2010 Dec 17;1(2):147–57.
- 28. Nakanishi N, Takashima T, Oto J. Muscle atrophy in critically ill patients: a review of its cause, evaluation, and prevention. The Journal of Medical Investigation. 2020;67(1.2):1–10.
- 29. Latronico N, Herridge M, Hopkins RO, Angus D, Hart N, Hermans G, et al. The ICM research agenda on intensive care unit-acquired weakness. Intensive Care Med. 2017 Sep 13;43(9):1270–81.
- 30. Price DR, Mikkelsen ME, Umscheid CA, Armstrong EJ. Neuromuscular Blocking Agents and Neuromuscular Dysfunction Acquired in Critical Illness: A Systematic Review and Meta-Analysis. Crit Care Med. 2016 Nov;44(11):2070–8.
- 31. Kanova M, Kohout P. Molecular Mechanisms Underlying Intensive Care Unit-Acquired Weakness and Sarcopenia. Int J Mol Sci. 2022 Jul 29;23(15):8396.
- 32. Bloch S, Polkey MI, Griffiths M, Kemp P. Molecular mechanisms of intensive care unit-acquired weakness. European Respiratory Journal. 2012 Apr;39(4):1000–11.
- 33. Friedrich O, Reid MB, Van den Berghe G, Vanhorebeek I, Hermans G, Rich MM, et al. The Sick and the Weak: Neuropathies/Myopathies in the Critically III. Physiol Rev. 2015 Jul;95(3):1025–109.
- 34. Vanhorebeek I, Latronico N, Van den Berghe G. ICU-acquired weakness. Intensive Care Med. 2020 Apr 19;46(4):637–53.
- 35. Piva S, Fagoni N, Latronico N. Intensive care unit–acquired weakness: unanswered questions and targets for future research. F1000Res. 2019 Apr 17;8:508.
- 36. Stevens RD, Marshall SA, Cornblath DR, Hoke A, Needham DM, de Jonghe B, et al. A framework for diagnosing and classifying intensive care unit-acquired weakness. Crit Care Med. 2009 Oct;37:S299–308.
- 37. Formenti P, Umbrello M, Coppola S, Froio S, Chiumello D. Clinical review: peripheral muscular ultrasound in the ICU. Ann Intensive Care. 2019 Dec 17;9(1):57.
- 38. Lad H, Saumur TM, Herridge MS, dos Santos CC, Mathur S, Batt J, et al. Intensive Care Unit-Acquired Weakness: Not Just Another Muscle Atrophying Condition. Int J Mol Sci. 2020 Oct 22;21(21):7840.
- 39. Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, et al. Acute Skeletal Muscle Wasting in Critical Illness. JAMA. 2013 Oct 16;310(15):1591.
- Hickmann CE, Castanares-Zapatero D, Deldicque L, Van den Bergh P, Caty G, Robert A, et al. Impact of Very Early Physical Therapy During Septic Shock on Skeletal Muscle: A Randomized Controlled Trial. Crit Care Med. 2018 Sep;46(9):1436–43.

- 41. Elkalawy H, Sekhar P, Abosena W. Early detection and assessment of intensive care unit-acquired weakness: a comprehensive review. Acute and Critical Care. 2023 Nov 30;38(4):409–24.
- 42. Weber-Carstens S, Schneider J, Wollersheim T, Assmann A, Bierbrauer J, Marg A, et al. Critical Illness Myopathy and GLUT4. Am J Respir Crit Care Med. 2013 Feb 15:187(4):387–96.
- 43. Appleton RT, Kinsella J, Quasim T. The incidence of intensive care unit-acquired weakness syndromes: A systematic review. J Intensive Care Soc. 2015 May 18;16(2):126–36.
- 44. Batt J, Mathur S, Katzberg HD. Mechanism of ICU-acquired weakness: muscle contractility in critical illness. Intensive Care Med. 2017 Apr 3;43(4):584–6.
- 45. Sidiras G, Patsaki I, Karatzanos E, Dakoutrou M, Kouvarakos A, Mitsiou G, et al. Long term follow-up of quality of life and functional ability in patients with ICU acquired Weakness A post hoc analysis. J Crit Care. 2019 Oct;53:223–30.
- 46. Castro-Ávila AC, Merino-Osorio C, González-Seguel F, Camus-Molina A, Leppe J. Impact on Mental, Physical and Cognitive functioning of a Critical care sTay during the COVID-19 pandemic (IMPACCT COVID-19): protocol for a prospective, multicentre, mixed-methods cohort study. BMJ Open. 2021 Sep 8;11(9):e053610.
- 47. Batt J, Herridge MS, dos Santos CC. From skeletal muscle weakness to functional outcomes following critical illness: a translational biology perspective. Thorax. 2019 Nov;74(11):1091–8.
- 48. Batt J, dos Santos CC, Cameron JI, Herridge MS. Intensive Care Unit–acquired Weakness. Am J Respir Crit Care Med. 2013 Feb 1;187(3):238–46.
- 49. dos Santos C, Hussain SNA, Mathur S, Picard M, Herridge M, Correa J, et al. Mechanisms of Chronic Muscle Wasting and Dysfunction after an Intensive Care Unit Stay. A Pilot Study. Am J Respir Crit Care Med. 2016 Oct 1;194(7):821–30.
- 50. Gunst J, Derese I, Aertgeerts A, Ververs EJ, Wauters A, Van den Berghe G, et al. Insufficient Autophagy Contributes to Mitochondrial Dysfunction, Organ Failure, and Adverse Outcome in an Animal Model of Critical Illness\*. Crit Care Med. 2013 Jan;41(1):182–94.
- 51. Banduseela VC, Chen YW, Kultima HG, Norman HS, Aare S, Radell P, et al. Impaired autophagy, chaperone expression, and protein synthesis in response to critical illness interventions in porcine skeletal muscle. Physiol Genomics. 2013 Jun 15;45(12):477–86.
- 52. Banduseela VC, Ochala J, Chen YW, Göransson H, Norman H, Radell P, et al. Gene expression and muscle fiber function in a porcine ICU model. Physiol Genomics. 2009 Nov;39(3):141–59.
- 53. Dos Santos CC, Batt J. ICU-acquired weakness. Curr Opin Crit Care. 2012 Oct;18(5):509–17.
- 54. Tuttle CSL, Thang LAN, Maier AB. Markers of inflammation and their association with muscle strength and mass: A systematic review and meta-analysis. Ageing Res Rev. 2020 Dec;64:101185.
- 55. Haberecht-Müller S, Krüger E, Fielitz J. Out of Control: The Role of the Ubiquitin Proteasome System in Skeletal Muscle during Inflammation. Biomolecules. 2021 Sep 8;11(9):1327.
- 56. Dinarello CA. Interleukin-1β. Crit Care Med. 2005 Dec;33(Suppl):S460–2.
- 57. Blevins HM, Xu Y, Biby S, Zhang S. The NLRP3 Inflammasome Pathway: A Review of Mechanisms and Inhibitors for the Treatment of Inflammatory Diseases. Front Aging Neurosci. 2022 Jun 10;14.
- 58. Ralston JC, Lyons CL, Kennedy EB, Kirwan AM, Roche HM. Fatty Acids and NLRP3 Inflammasome–Mediated Inflammation in Metabolic Tissues. Annu Rev Nutr. 2017 Aug 21;37(1):77–102.
- 59. Sayed RK, Fernández-Ortiz M, Fernández-Martínez J, Aranda Martínez P, Guerra-Librero A, Rodríguez-Santana C, et al. The Impact of Melatonin and NLRP3 Inflammasome on the Expression of microRNAs in Aged Muscle. Antioxidants. 2021 Mar 27;10(4):524.

- 60. Jorquera G, Russell J, Monsalves-Álvarez M, Cruz G, Valladares-Ide D, Basualto-Alarcón C, et al. NLRP3 Inflammasome: Potential Role in Obesity Related Low-Grade Inflammation and Insulin Resistance in Skeletal Muscle. Int J Mol Sci. 2021 Mar 23;22(6):3254.
- 61. Moreno-García L, Miana-Mena FJ, Moreno-Martínez L, de la Torre M, Lunetta C, Tarlarini C, et al. Inflammasome in ALS Skeletal Muscle: NLRP3 as a Potential Biomarker. Int J Mol Sci. 2021 Mar 3;22(5):2523.
- 62. Sayed RK, Fernández-Ortiz M, Fernández-Martínez J, Aranda Martínez P, Guerra-Librero A, Rodríguez-Santana C, et al. The Impact of Melatonin and NLRP3 Inflammasome on the Expression of microRNAs in Aged Muscle. Antioxidants. 2021 Mar 27;10(4):524.
- 63. Antuña E, Potes Y, Baena-Huerta FJ, Cachán-Vega C, Menéndez-Coto N, Álvarez Darriba E, et al. NLRP3 Contributes to Sarcopenia Associated to Dependency Recapitulating Inflammatory-Associated Muscle Degeneration. Int J Mol Sci. 2024 Jan 24;25(3):1439.
- 64. McBride MJ, Foley KP, D'Souza DM, Li YE, Lau TC, Hawke TJ, et al. The NLRP3 inflammasome contributes to sarcopenia and lower muscle glycolytic potential in old mice. American Journal of Physiology-Endocrinology and Metabolism. 2017 Aug 1;313(2):E222–32.
- 65. Eggelbusch M, Shi A, Broeksma BC, Vázquez-Cruz M, Soares MN, de Wit GMJ, et al. The NLRP3 inflammasome contributes to inflammation-induced morphological and metabolic alterations in skeletal muscle. J Cachexia Sarcopenia Muscle. 2022 Dec 17;13(6):3048–61.
- 66. Llano-Diez M, Fury W, Okamoto H, Bai Y, Gromada J, Larsson L. RNA-sequencing reveals altered skeletal muscle contraction, E3 ligases, autophagy, apoptosis, and chaperone expression in patients with critical illness myopathy. Skelet Muscle. 2019 Dec 16;9(1):9.
- 67. Walsh CJ, Batt J, Herridge MS, Mathur S, Bader GD, Hu P, et al. Transcriptomic analysis reveals abnormal muscle repair and remodeling in survivors of critical illness with sustained weakness. Sci Rep. 2016 Jul 14;6(1):29334.
- 68. Huang N, Kny M, Riediger F, Busch K, Schmidt S, Luft FC, et al. Deletion of Nlrp3 protects from inflammation-induced skeletal muscle atrophy. Intensive Care Med Exp. 2017 Dec 17;5(1):3.
- 69. You Z, Huang X, Xiang Y, Dai J, Xu L, Jiang J, et al. Ablation of NLRP3 inflammasome attenuates muscle atrophy via inhibiting pyroptosis, proteolysis and apoptosis following denervation. Theranostics. 2023;13(1):374–90.
- 70. Hussain SNA, Mofarrahi M, Sigala I, Kim HC, Vassilakopoulos T, Maltais F, et al. Mechanical Ventilation–induced Diaphragm Disuse in Humans Triggers Autophagy. Am J Respir Crit Care Med. 2010 Dec 1;182(11):1377–86.
- 71. Constantin D, McCullough J, Mahajan RP, Greenhaff PL. Novel events in the molecular regulation of muscle mass in critically ill patients. J Physiol. 2011 Aug 1;589(15):3883–95.
- 72. Klaude M, Mori M, Tjäder I, Gustafsson T, Wernerman J, Rooyackers O. Protein metabolism and gene expression in skeletal muscle of critically ill patients with sepsis. Clin Sci. 2012 Feb 1;122(3):133–42.
- 73. Schmidt F, Kny M, Zhu X, Wollersheim T, Persicke K, Langhans C, et al. The E3 ubiquitin ligase TRIM62 and inflammation-induced skeletal muscle atrophy. Crit Care. 2014 Oct 29;18(5):545.
- 74. Wray CJ, Mammen JMV, Hershko DD, Hasselgren PO. Sepsis upregulates the gene expression of multiple ubiquitin ligases in skeletal muscle. Int J Biochem Cell Biol. 2003 May;35(5):698–705.
- 75. Ochala J, Gustafson AM, Diez ML, Renaud G, Li M, Aare S, et al. Preferential skeletal muscle myosin loss in response to mechanical silencing in a novel rat intensive care unit model: underlying mechanisms. J Physiol. 2011 Apr;589(8):2007–26.
- 76. Corpeno Kalamgi R, Salah H, Gastaldello S, Martinez-Redondo V, Ruas JL, Fury W, et al. Mechano-signalling pathways in an experimental intensive critical illness myopathy model. J Physiol. 2016 Aug 1;594(15):4371–88.

- 77. Salah H, Fury W, Gromada J, Bai Y, Tchkonia T, Kirkland JL, et al. Muscle-specific differences in expression and phosphorylation of the Janus kinase 2/Signal Transducer and Activator of Transcription 3 following long-term mechanical ventilation and immobilization in rats. Acta Physiologica. 2018 Mar 30;222(3).
- 78. Cacciani N, Salah H, Li M, Akkad H, Backeus A, Hedstrom Y, et al. Chaperone coinducer BGP-15 mitigates early contractile dysfunction of the soleus muscle in a rat ICU model. Acta Physiologica. 2020 May 18;229(1).
- 79. Ozdemir M, Bomkamp MP, Hyatt HW, Smuder AJ, Powers SK. Intensive Care Unit Acquired Weakness Is Associated with Rapid Changes to Skeletal Muscle Proteostasis. Cells. 2022 Dec 11;11(24):4005.
- 80. Renaud G, Llano-Diez M, Ravara B, Gorza L, Feng HZ, Jin JP, et al. Sparing of muscle mass and function by passive loading in an experimental intensive care unit model. J Physiol. 2013 Mar;591(5):1385–402.
- 81. Zanders L, Kny M, Hahn A, Schmidt S, Wundersitz S, Todiras M, et al. Sepsis induces interleukin 6, gp130/JAK2/STAT3, and muscle wasting. J Cachexia Sarcopenia Muscle. 2022 Feb 24;13(1):713–27.
- 82. Van Dyck L, Güiza F, Derese I, Pauwels L, Casaer MP, Hermans G, et al. DNA methylation alterations in muscle of critically ill patients. J Cachexia Sarcopenia Muscle. 2022 Jun 11;13(3):1731–40.
- 83. Klaude M, Fredriksson K, Tjäder I, Hammarqvist F, Ahlman B, Rooyackers O, et al. Proteasome proteolytic activity in skeletal muscle is increased in patients with sepsis. Clin Sci. 2007 May 1;112(9):499–506.
- 84. Liu Y, Wang D, Li T, Yang F, Li Z, Bai X, et al. The role of NLRP3 inflammasome in inflammation-related skeletal muscle atrophy. Front Immunol. 2022 Nov 3;13.
- 85. Swanson K V., Deng M, Ting JPY. The NLRP3 inflammasome: molecular activation and regulation to therapeutics. Nat Rev Immunol. 2019 Aug 29;19(8):477–89.
- 86. Chen C, Xu P. Activation and Pharmacological Regulation of Inflammasomes. Biomolecules. 2022 Jul 20;12(7):1005.
- 87. Yang T, Li Z, Jiang L, Wang Y, Xi X. Risk factors for intensive care unit-acquired weakness: A systematic review and meta-analysis. Acta Neurol Scand. 2018 Aug;138(2):104–14.
- 88. Puthucheary ZA, Astin R, Mcphail MJW, Saeed S, Pasha Y, Bear DE, et al. Metabolic phenotype of skeletal muscle in early critical illness. Thorax. 2018 Oct;73(10):926–35.
- 89. Zhao K, Li X, Zhang M, Tong F, Chen H, Wang X, et al. microRNA-181a Promotes Mitochondrial Dysfunction and Inflammatory Reaction in a Rat Model of Intensive Care Unit-Acquired Weakness by Inhibiting IGFBP5 Expression. J Neuropathol Exp Neurol. 2022 Jun 20;81(7):553–64.
- 90. Cacciani N, Skärlén Å, Wen Y, Zhang X, Addinsall AB, Llano-Diez M, et al. A prospective clinical study on the mechanisms underlying critical illness myopathy—A time-course approach. J Cachexia Sarcopenia Muscle. 2022 Dec 12;13(6):2669–82.
- 91. Kelley N, Jeltema D, Duan Y, He Y. The NLRP3 Inflammasome: An Overview of Mechanisms of Activation and Regulation. Int J Mol Sci. 2019 Jul 6;20(13):3328.
- 92. Xu M, Wang L, Wang M, Wang H, Zhang H, Chen Y, et al. Mitochondrial ROS and NLRP3 inflammasome in acute ozone-induced murine model of airway inflammation and bronchial hyperresponsiveness. Free Radic Res. 2019 Jul 3;53(7):780–90.
- 93. Hou Y, Wang Q, Han B, Chen Y, Qiao X, Wang L. CD36 promotes NLRP3 inflammasome activation via the mtROS pathway in renal tubular epithelial cells of diabetic kidneys. Cell Death Dis. 2021 May 21;12(6):523.
- 94. Sho T, Xu J. Role and mechanism of ROS scavengers in alleviating NLRP3-mediated inflammation. Biotechnol Appl Biochem. 2019 Jan 25;66(1):4–13.
- 95. Carré JE, Orban JC, Re L, Felsmann K, Iffert W, Bauer M, et al. Survival in Critical Illness Is Associated with Early Activation of Mitochondrial Biogenesis. Am J Respir Crit Care Med. 2010 Sep 15;182(6):745–51.
- 96. Salah H, Li M, Cacciani N, Gastaldello S, Ogilvie H, Akkad H, et al. The chaperone coinducer BGP-15 alleviates ventilation-induced diaphragm dysfunction. Sci Transl Med. 2016 Aug 3;8(350).

- 97. Owen AM, Patel SP, Smith JD, Balasuriya BK, Mori SF, Hawk GS, et al. Chronic muscle weakness and mitochondrial dysfunction in the absence of sustained atrophy in a preclinical sepsis model. Elife. 2019 Dec 3;8.
- 98. Mofarrahi M, Sigala I, Guo Y, Godin R, Davis EC, Petrof B, et al. Autophagy and Skeletal Muscles in Sepsis. PLoS One. 2012 Oct 9;7(10):e47265.
- 99. Fredriksson K, Hammarqvist F, Strigård K, Hultenby K, Ljungqvist O, Wernerman J, et al. Derangements in mitochondrial metabolism in intercostal and leg muscle of critically ill patients with sepsis-induced multiple organ failure. American Journal of Physiology-Endocrinology and Metabolism. 2006 Nov;291(5):E1044–50.
- 100. Picard M, Jung B, Liang F, Azuelos I, Hussain S, Goldberg P, et al. Mitochondrial Dysfunction and Lipid Accumulation in the Human Diaphragm during Mechanical Ventilation. Am J Respir Crit Care Med. 2012 Dec 1;186(11):1140–9.
- 101. Fredriksson K, Tjäder I, Keller P, Petrovic N, Ahlman B, Schéele C, et al. Dysregulation of Mitochondrial Dynamics and the Muscle Transcriptome in ICU Patients Suffering from Sepsis Induced Multiple Organ Failure. PLoS One. 2008 Nov 10;3(11):e3686.
- 102. Puthucheary ZA, Astin R, Mcphail MJW, Saeed S, Pasha Y, Bear DE, et al. Metabolic phenotype of skeletal muscle in early critical illness. Thorax. 2018 Oct;73(10):926–35.
- 103. Rocheteau P, Chatre L, Briand D, Mebarki M, Jouvion G, Bardon J, et al. Sepsis induces long-term metabolic and mitochondrial muscle stem cell dysfunction amenable by mesenchymal stem cell therapy. Nat Commun. 2015 Dec 15;6(1):10145.
- 104. Vanhorebeek I, Gunst J, Derde S, Derese I, Boussemaere M, Güiza F, et al. Insufficient Activation of Autophagy Allows Cellular Damage to Accumulate in Critically III Patients. J Clin Endocrinol Metab. 2011 Apr 1;96(4):E633–45.
- 105. Brealey D, Brand M, Hargreaves I, Heales S, Land J, Smolenski R, et al. Association between mitochondrial dysfunction and severity and outcome of septic shock. The Lancet. 2002 Jul;360(9328):219–23.
- 106. Jiroutková K, Krajčová A, Ziak J, Fric M, Waldauf P, Džupa V, et al. Mitochondrial function in skeletal muscle of patients with protracted critical illness and ICU-acquired weakness. Crit Care. 2015 Dec 6;19(1):448.
- 107. Tang H, Smith IJ, Hussain SNA, Goldberg P, Lee M, Sugiarto S, et al. The JAK-STAT Pathway Is Critical in Ventilator-Induced Diaphragm Dysfunction. Molecular Medicine. 2014 Jan 30;20(1):579–89.
- 108. Thomas D, Maes K, Agten A, Heunks L, Dekhuijzen R, Decramer M, et al. Time course of diaphragm function recovery after controlled mechanical ventilation in rats. J Appl Physiol. 2013 Sep 15;115(6):775–84.
- 109. Llano-Diez M, Renaud G, Andersson M, Marrero H, Cacciani N, Engquist H, et al. Mechanisms underlying ICU muscle wasting and effects of passive mechanical loading. Crit Care. 2012;16(1):R209.
- 110. Chevriaux A, Pilot T, Derangère V, Simonin H, Martine P, Chalmin F, et al. Cathepsin B Is Required for NLRP3 Inflammasome Activation in Macrophages, Through NLRP3 Interaction. Front Cell Dev Biol. 2020 Mar 31;8.
- 111. Doiron KA, Hoffmann TC, Beller EM. Early intervention (mobilization or active exercise) for critically ill adults in the intensive care unit. Cochrane Database of Systematic Reviews. 2018 Mar 27;2018(12).
- 112. Reid JC, Unger J, McCaskell D, Childerhose L, Zorko DJ, Kho ME. Physical rehabilitation interventions in the intensive care unit: a scoping review of 117 studies. J Intensive Care. 2018 Dec 7;6(1):80.
- 113. Tipping CJ, Harrold M, Holland A, Romero L, Nisbet T, Hodgson CL. The effects of active mobilisation and rehabilitation in ICU on mortality and function: a systematic review. Intensive Care Med. 2017 Feb 18;43(2):171–83.
- 114. Fuke R, Hifumi T, Kondo Y, Hatakeyama J, Takei T, Yamakawa K, et al. Early rehabilitation to prevent postintensive care syndrome in patients with critical illness: a systematic review and meta-analysis. BMJ Open. 2018 May 5;8(5):e019998.
- 115. Zhang L, Hu W, Cai Z, Liu J, Wu J, Deng Y, et al. Early mobilization of critically ill patients in the intensive care unit: A systematic review and meta-analysis. PLoS One. 2019 Oct 3;14(10):e0223185.

- 116. Heidegger CP, Berger MM, Graf S, Zingg W, Darmon P, Costanza MC, et al. Optimisation of energy provision with supplemental parenteral nutrition in critically ill patients: a randomised controlled clinical trial. The Lancet. 2013 Feb;381(9864):385–93.
- 117. Kim JY, Kwon YG, Kim YM. The stress-responsive protein REDD1 and its pathophysiological functions. Exp Mol Med. 2023 Sep 1;55(9):1933–44.
- 118. Zhao R. Exercise mimetics: a novel strategy to combat neuroinflammation and Alzheimer's disease. J Neuroinflammation. 2024 Feb 2;21(1):40.
- 119. Scheffer D da L, Latini A. Exercise-induced immune system response: Anti-inflammatory status on peripheral and central organs. Biochimica et Biophysica Acta (BBA) Molecular Basis of Disease. 2020 Oct;1866(10):165823.
- 120. Wang J, Liu S, Li G, Xiao J. Exercise Regulates the Immune System. In 2020. p. 395–408.
- 121. Ringseis R, Eder K, Mooren FC, Krüger K. Metabolic signals and innate immune activation in obesity and exercise. Exerc Immunol Rev. 2015;21:58–68.
- 122. Courel-Ibáñez J, Vetrovsky T, Růžičková N, Marañón C, Durkalec-Michalski K, Tomcik M, et al. Integrative non-pharmacological care for individuals at risk of rheumatoid arthritis. Rheumatol Int. 2024 Jan 5;44(3):413–23.
- 123. Calabrese L, Nieman DC. Exercise, infection and rheumatic diseases: what do we know? RMD Open. 2021 May;7(2):e001644.
- 124. Safdar NZ, Alobaid AM, Hopkins M, Dempsey PC, Pearson SM, Kietsiriroje N, et al. Short, frequent, light-intensity walking activity improves postprandial vascular-inflammatory biomarkers in people with type 1 diabetes: The <scp>SIT-LESS</scp>randomized controlled trial. Diabetes Obes Metab. 2024 Jun;26(6):2439–45.
- 125. Pairo Z, Parnow A, Sari Aslani P, Mohammadi P, Mirzaeei S, Mohr M. Exercise training reduces systemic inflammation and improves general health status in female migraineurs: a randomised controlled trail. Eur J Appl Physiol. 2024 May 3;124(5):1397–408.
- 126. Valero-Breton M, Valladares-Ide D, Álvarez C, Peñailillo RS, Peñailillo L. Changes in Blood Markers of Oxidative Stress, Inflammation and Cardiometabolic Patients with COPD after Eccentric and Concentric Cycling Training. Nutrients. 2023 Feb 11;15(4):908.
- 127. Gao K, Su Z, Meng J, Yao Y, Li L, Su Y, et al. Effect of Exercise Training on Some Anti-Inflammatory Adipokines, High Sensitivity C-Reactive Protein, and Clinical Outcomes in Sedentary Adults With Metabolic Syndrome. Biol Res Nurs. 2024 Jan 14;26(1):125–38.
- 128. Son WH, Park HT, Jeon BH, Ha MS. Moderate intensity walking exercises reduce the body mass index and vascular inflammatory factors in postmenopausal women with obesity: a randomized controlled trial. Sci Rep. 2023 Nov 17;13(1):20172.
- 129. Hu J, Wang Y, Ji X, Zhang Y, Li K, Huang F. Non-Pharmacological Strategies for Managing Sarcopenia in Chronic Diseases. Clin Interv Aging. 2024 May; Volume 19:827–41.
- 130. Ringleb M, Javelle F, Haunhorst S, Bloch W, Fennen L, Baumgart S, et al. Beyond muscles: Investigating immunoregulatory myokines in acute resistance exercise A systematic review and meta-analysis. The FASEB Journal. 2024 Apr 15;38(7).
- 131. Ding Y, Xu X. Anti-inflammatory effect of exercise training through reducing inflammasome activation-related inflammatory cytokine levels in overweight/obese populations: A systematic review and meta-analysis. Complement Ther Clin Pract. 2022 Nov:49:101656.
- 132. Luo B, Xiang D, Ji X, Chen X, Li R, Zhang S, et al. The anti-inflammatory effects of exercise on autoimmune diseases: A 20-year systematic review. J Sport Health Sci. 2024 May;13(3):353–67.
- 133. Mejías-Peña Y, Estébanez B, Rodriguez-Miguelez P, Fernandez-Gonzalo R, Almar M, de Paz JA, et al. Impact of resistance training on the autophagy-inflammation-apoptosis crosstalk in elderly subjects. Aging. 2017 Feb 2;9(2):408–18.
- 134. Wang W, Lv Z, Gao J, Liu M, Wang Y, Tang C, et al. Treadmill exercise alleviates neuronal damage by suppressing NLRP3 inflammasome and microglial activation in

- the MPTP mouse model of Parkinson's disease. Brain Res Bull. 2021 Sep;174:349–58
- 135. Li C, Xu X, Wang Z, Wang Y, Luo L, Cheng J, et al. Exercise ameliorates post-stroke depression by inhibiting PTEN elevation-mediated upregulation of TLR4/NF-κB/NLRP3 signaling in mice. Brain Res. 2020 Jun;1736:146777.
- 136. Zhang Y, Liu Y, Bi X, Hu C, Ding F, Ding W. Therapeutic Approaches in Mitochondrial Dysfunction, Inflammation, and Autophagy in Uremic Cachexia: Role of Aerobic Exercise. Mediators Inflamm. 2019 Aug 18;2019:1–11.
- 137. Grace PM, Fabisiak TJ, Green-Fulgham SM, Anderson ND, Strand KA, Kwilasz AJ, et al. Prior voluntary wheel running attenuates neuropathic pain. Pain. 2016 Sep;157(9):2012–23.
- 138. Pelaia TM, Shojaei M, McLean AS. The Role of Transcriptomics in Redefining Critical Illness. Crit Care. 2023 Mar 21;27(1):89.
- 139. Montgomery SB, Bernstein JA, Wheeler MT. Toward transcriptomics as a primary tool for rare disease investigation. Cold Spring Harb Mol Case Stud. 2022 Feb;8(2).
- 140. Tsakiroglou M, Evans A, Pirmohamed M. Leveraging transcriptomics for precision diagnosis: Lessons learned from cancer and sepsis. Front Genet. 2023 Mar 10;14.
- 141. Langhans C, Weber-Carstens S, Schmidt F, Hamati J, Kny M, Zhu X, et al. Inflammation-Induced Acute Phase Response in Skeletal Muscle and Critical Illness Myopathy. PLoS One. 2014 Mar 20;9(3):e92048.
- 142. Llano-Diez M, Gustafson AM, Olsson C, Goransson H, Larsson L. Muscle wasting and the temporal gene expression pattern in a novel rat intensive care unit model. BMC Genomics. 2011 Dec 13;12(1):602.
- 143. Ju M, Bi J, Wei Q, Jiang L, Guan Q, Zhang M, et al. Pan-cancer analysis of NLRP3 inflammasome with potential implications in prognosis and immunotherapy in human cancer. Brief Bioinform. 2021 Jul 20;22(4).
- 144. Wollersheim T, Woehlecke J, Krebs M, Hamati J, Lodka D, Luther-Schroeder A, et al. Dynamics of myosin degradation in intensive care unit-acquired weakness during severe critical illness. Intensive Care Med. 2014 Apr 15;40(4):528–38.
- 145. Hough CL, Lieu BK, Caldwell ES. Manual muscle strength testing of critically ill patients: feasibility and interobserver agreement. Crit Care. 2011;15(1):R43.
- 146. Nickels MR, Aitken LM, Barnett AG, Walsham J, King S, Gale NE, et al. Effect of inbed cycling on acute muscle wasting in critically ill adults: A randomised clinical trial. J Crit Care. 2020 Oct;59:86–93.
- 147. Kho ME, Berney S, Pastva AM, Kelly L, Reid JC, Burns KEA, et al. Early In-Bed Cycle Ergometry in Mechanically Ventilated Patients. NEJM Evidence. 2024 Jun 25;3(7).
- 148. Nickels MR, Aitken LM, Walsham J, Barnett AG, McPhail SM. Critical Care Cycling Study (CYCLIST) trial protocol: a randomised controlled trial of usual care plus additional in-bed cycling sessions versus usual care in the critically ill. BMJ Open. 2017 Oct 22;7(10):e017393.
- 149. Hodgson CL, Stiller K, Needham DM, Tipping CJ, Harrold M, Baldwin CE, et al. Expert consensus and recommendations on safety criteria for active mobilization of mechanically ventilated critically ill adults. Crit Care. 2014 Dec 4;18(6):658.
- 150. Crawford AM, Shiferaw AA, Ntambwe P, Milan AO, Khalid K, Rubio R, et al. Global critical care: a call to action. Crit Care. 2023 Jan 20;27(1):28.
- 151. Garros RF, Paul R, Connolly M, Lewis A, Garfield BE, Natanek SA, et al. MicroRNA-542 Promotes Mitochondrial Dysfunction and SMAD Activity and Is Elevated in Intensive Care Unit–acquired Weakness. Am J Respir Crit Care Med. 2017 Dec 1;196(11):1422–33.
- 152. Pietrangelo T, Perni S, Di Tano G, Fanó-Illic G, Franzini-Armstrong C. A method for the ultrastructural preservation of tiny percutaneous needle biopsy material from skeletal muscle. Int J Mol Med. 2013 Oct;32(4):965–70.
- 153. Turan Z, Topaloglu M, Ozyemisci Taskiran O. Medical Research Council-sumscore: a tool for evaluating muscle weakness in patients with post-intensive care syndrome. Crit Care. 2020 Dec 18;24(1):562.
- 154. Mittal S, Hadda V, Khilnani GC, Dhunguna A, Khan MA. Intra- and Inter-Observer Reliability of Quadriceps Muscle Thickness Measured with Bedside Ultrasonography

- by Critical Care Physicians. Indian Journal of Critical Care Medicine. 2017 Jul:21(7):448–52.
- 155. Di Matteo A, Moscioni E, Lommano MG, Cipolletta E, Smerilli G, Farah S, et al. Reliability assessment of ultrasound muscle echogenicity in patients with rheumatic diseases: Results of a multicenter international web-based study. Front Med (Lausanne). 2023 Jan 17;9.
- 156. Pardo E, El Behi H, Boizeau P, Verdonk F, Alberti C, Lescot T. Reliability of ultrasound measurements of quadriceps muscle thickness in critically ill patients. BMC Anesthesiol. 2018 Dec 27;18(1):205.
- 157. Karapınar M, Atilla Ayyıldız V, Ünal M, Fırat T. Ultrasound imaging of quadriceps muscle in patients with knee osteoarthritis: The test-retest and inter-rater reliability and concurrent validity of echo intensity measurement. Musculoskelet Sci Pract. 2021 Dec;56:102453.
- 158. González-Seguel F, Camus-Molina A, Cárcamo M, Hiser S, Needham DM, Leppe J. Inter-observer reliability of trained physiotherapists on the Functional Status Score for the Intensive Care Unit Chilean-Spanish version. Physiother Theory Pract. 2022 Feb 1;38(2):365–71.
- 159. Mahoney DJ, Carey K, Fu MH, Snow R, Cameron-Smith D, Parise G, et al. Real-time RT-PCR analysis of housekeeping genes in human skeletal muscle following acute exercise. Physiol Genomics. 2004 Jul 8;18(2):226–31.
- 160. Moïsi L, Mino JC, Guidet B, Vallet H. Frailty assessment in critically ill older adults: a narrative review. Ann Intensive Care. 2024 Jun 18;14(1):93.
- 161. Tipping CJ, Young PJ, Romero L, Saxena MK, Dulhunty J, Hodgson CL. A systematic review of measurements of physical function in critically ill adults. Crit Care Resusc. 2012 Dec;14(4):302–11.
- 162. Caceres-Parra C, González-Seguel F, Merino-Osorio C, Adasme R. National survey of changes in the practices of critical care physiotherapists during the COVID-19 pandemic in Chile: DeKUCI COVID-19 Study. Santiago; 2021.
- 163. de Letter MACJ, Schmitz PIM, Visser LH, Verheul FAM, Schellens RLLA, Op de Coul DAW, et al. Risk factors for the development of polyneuropathy and myopathy in critically ill patients. Crit Care Med. 2001 Dec;29(12):2281–6.
- 164. Kho MĚ, Molloy AJ, Clarke F, Herridge MS, Koo KKY, Rudkowski J, et al. CYCLE pilot: a protocol for a pilot randomised study of early cycle ergometry versus routine physiotherapy in mechanically ventilated patients. BMJ Open. 2016 Apr 8;6(4):e011659.
- 165. Raithatha A, Ashraghi MR, Lord C, Limback-Stanic C, Viegas S, Amiras D. Ultrasound-guided muscle biopsy: a practical alternative for investigation of myopathy. Skeletal Radiol. 2020 Nov 9;49(11):1855–9.
- 166. Messina A, Robba C, Bertuetti R, Biasucci D, Corradi F, Mojoli F, et al. Head to toe ultrasound: a narrative review of experts' recommendations of methodological approaches. Journal of Anesthesia, Analgesia and Critical Care. 2022 Oct 21;2(1):44.
- 167. Chasset F, Soria A, Moguelet P, Mathian A, Auger Y, Francès C, et al. Contact dermatitis due to ultrasound gel: A case report and published work review. J Dermatol. 2016 Mar 8;43(3):318–20.
- 168. Cacciapuoti S, Masarà A, Fabbrocini G, Patruno C. Contact Urticaria to Ultrasound Gel: A Case Report. Dermatitis. 2018 Mar;29(2):93–93.
- 169. Martínez Antón MD, Jáuregui I, Galán C, Sánchez de Vicente J, Segurola A, Seras Y, et al. Two cases of allergic contact dermatitis to different elements in identical ultrasound gels. Contact Dermatitis. 2021 Oct 25;85(4):477–8.
- 170. Villa A, Venegoni M, Tiso B. Cases of contact dermatitis caused by ultrasonographic gel. Journal of Ultrasound in Medicine. 1998 Aug;17(8):530–530.
- 171. KESSLER J, SCHAFHALTERZOPPOTH I, GRAY A. Allergic Contact Dermatitis Caused by Ultrasonic Gel. Reg Anesth Pain Med. 2006 Sep;31(5):480–1.
- 172. Chasset F, Soria A, Moguelet P, Mathian A, Auger Y, Francès C, et al. Contact dermatitis due to ultrasound gel: A case report and published work review. J Dermatol. 2016 Mar 8;43(3):318–20.

- 173. Neves JM, Barreto G, Boobis L, Harris R, Roschel H, Tricoli V, et al. Incidence of adverse events associated with percutaneous muscular biopsy among healthy and diseased subjects. Scand J Med Sci Sports. 2012 Apr 10;22(2):175–8.
- 174. Ekblom B. The muscle biopsy technique. Historical and methodological considerations. Scand J Med Sci Sports. 2017 May 29;27(5):458–61.
- 175. Cerino M, González-Hormazábal P, Abaji M, Courrier S, Puppo F, Mathieu Y, et al. Genetic Profile of Patients with Limb-Girdle Muscle Weakness in the Chilean Population. Genes (Basel). 2022 Jun 16;13(6):1076.
- 176. Américo-Da-Silva L, Aguilera J, Quinteros-Waltemath O, Sánchez-Aguilera P, Russell J, Cadagan C, et al. Activation of the NLRP3 Inflammasome Increases the IL-1β Level and Decreases GLUT4 Translocation in Skeletal Muscle during Insulin Resistance. Int J Mol Sci. 2021 Sep 23;22(19):10212.
- 177. Monsalves-Álvarez M, Solis-Soto MT, Burrone MS, Candia AA, Jofré-Saldía E, Espinoza G, et al. Community strategies for health promotion and prevention of chronic non-communicable diseases with a focus on physical activity and nutrition: the URO/FOCOS study protocol. Front Public Health. 2024 Jan 12;11.

# 10. Gantt Chart

| | | 24 | 2025 | | | | 2026 | |
|---|---|---|---|---|---|---|---|---|
| ACTIVIDAD | 3° | 4° | 1° | 2° | 3° - | 4° | 1° 2° | 3° 4° |
| OE1: Evaluar el efecto de la terapia física en la activación del inflamosoma NLRP3 en biopsias del vasto lateral de | | | | - | | | · | |
| pacientes con MPC, y comparar esta actividad con la de pacientes control. | | | | | | | | |
| Priming del inflamosoma NLRP3 - NLRP3, IL-1β e IL-18 mRNA - RT-qPCR | | | | | | | | |
| Priming del inflamosoma NLRP3 - p65S536/p65t - Western blot | | | | | | | | |
| Actividad del inflamosoma NLRP3 - Caspasa-1/pro-caspasa-1 IL-1β/pro-IL-1β GSDMD/NGSDMD - Western blot | $\perp$ | | | | | | | |
| Actividad del inflamosoma NLRP3. IL-1β - IL-18 - ELISA | | | | | | | | |
| Fact. ~ con ensamblaje I. NLRP3 - Estrés oxidativo - Dinitrofenol, Nitrotirosina - Western Blot | | | | | | | | |
| Fact. ~ con ensamblaje I. NLRP3 - Catepsina B - RT-qPCR/Western Blot | | | | | | | | |
| OE2: Evaluar el efecto de la terapia física sobre la atrofia muscular en biopsias de vasto lateral de pacientes con MPC, y relacionar estos resultados con la activación del inflamosoma NLRP3. | | | | | | | | |
| Diagnóstico molecular de la MPC - Razón Miosina/Actina - Western blot | | | | | | | | |
| Diagnóstico molecular de la MPC - Desorganización sarcomética - TEM | | | | | | | | |
| Atrofia muscular - IFI laminina | | | | | | | | |
| Atrogenes- MurF1, atrogina-1, MUSA1, TRIM62 y TRIM32 mRNA - RT-qPCR | | | | | | | | |
| OE3: Evaluar el efecto de la terapia física en el perfil de expresión génica de las vías de señalización involucradas en la atrofia del músculo esquelético en pacientes con MPC. | | | | | | | | |
| Ensayo de transcriptómica por Microarray | | | | | | | | |
| Análisis estadístico y bioinformático: DEG, GO | | | | | | | | |
| OE4: Analizar la asociación entre la expresión génica y los parámetros bioquímicos del músculo esquelético con | | | | | | | | |
| el diagnóstico clínico de la MPC. | + | 1 | | 1 1 | | - 1 | | |
| Análisis estadístico de la asociación entre los hallazgos bioquímicas del músculo y el diagnóstico clínico de la MPC. Otros | + | | | | | | | |
| Estandarización técnica: WB - RT-qPCR - Histología e IFI | | | | | Т | | | $\overline{}$ |
| Proyecto piloto Variabilidad inter-evaluador: MRC SS, FSS ICU, ecografía muscular y ecografía de nervio periférico | | | | | | | | <del> </del> |
| Examen de calificación | + | | | | | _ | _ | |
| Presentación provecto a Comité de Ética | + | | | | | _ | _ | |
| Presentación proyecto a SEREMI de Salud | + | + | | | | | | +- |
| Registro proyecto en ClinicalTrials | <del>† </del> | + | | | | | | <del> </del> |
| Escritura artículo científico - Protocolo | + | + | | | | - | | + |
| Diseño e incorporación plataforma REDCap | $\vdash$ | 1 | | | | $\dashv$ | | +- |
| Avance 1 | $\vdash$ | $\vdash$ | <u> </u> | | | | | $\vdash$ |
| Avance 2 | + | $\vdash$ | | H | - 1 | | + | |
| Escritura artículo científico | + | 1 | | H | | - | | |
| Escritura de tesis | + | 1 | 1 | | | -+ | | |
| Tesis final | $\vdash$ | $\vdash$ | | $\vdash$ | $\dashv$ | $\dashv$ | - | |
| resis iiriai | | | 1 | | | | | |



**Appendix 2. Ultrasound Evaluation Procedure** 

1. Muscle Ultrasound

Ultrasound assessments of the quadriceps muscle will be performed within the first 72 hours of ICU admission (Day 1) and again at Day 7. To identify the site for the transverse measurement, the patient will be placed in a supine position with the knee joint in a neutral resting position. A line will be drawn between the anterior superior iliac spine (ASIS) and the superior pole of the patella, and measurements will be taken at the junction between the middle and lower third of this line. At this measurement point, the thickness of the anterior quadriceps complex—including the rectus femoris (RF) and the vastus intermedius (VI)—as well as its cross-sectional area (CSA), will be assessed. Images will be acquired for echogenicity analysis using ImageJ software.

For longitudinal measurements, a point 5 cm lateral to the transverse measurement site will be marked, where the pennation angle will be evaluated. A linear transducer with a frequency range of 4 to 12 MHz (Sonosite<sup>™</sup>